CLINICAL TRIAL: NCT03547271
Title: Immunogenicity and Safety Study of an Investigational Quadrivalent Meningococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers in Europe
Brief Title: Immunogenicity and Safety Study of a Quadrivalent Meningococcal Conjugate Vaccine When Co-administered With Routine Pediatric Vaccines in Healthy Infants and Toddlers in Europe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET58; U1111-1183-6653 (Registry Identifier: ICTRP); MET58 (Other: Sanofi Identifier); 2017-004731-36 (EudraCT Number)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Meningococcal Infections
Keywords: Meningococcal meningitis; MenACYW conjugate vaccine; Quadrivalent meningococcal vaccine
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — 13-valent pneumococcal vaccine; 10-valent pneumococcal vaccine; PHiD-CV vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double blind for Groups 1 and 2 and open label for Groups 3 and 4 for meningococcal vaccines. Open-label for all concomitant routine vaccines.
  Modified double-blind: the participants parent / legally acceptable representative, the Investigator, and other study personnel remain unaware of the treatment assignments throughout the trial. An unblinded vaccine administrator will administer the appropriate vaccines but will not be involved in safety data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: MenACYW (Experimental): Participants received 3 doses of meningococcal polysaccharide (serogroups A, C, Y and W) tetanus toxoid [MenACYW conjugate vaccine] 0.5 milliliter (mL) as an intramuscular (IM) injection at dose 1: 2 months of age (MoA), dose 2: 4 MoA, and dose 3: 12 to 18 MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (combined diphtheria, tetanus, acellular pertussis, hepatitis B, inactivated poliovirus and haemophilus influenzae type b conjugate vaccine [DTaP-IPV-HB-Hib], the pneumococcal vaccine (pneumococcal conjugate vaccine [10-valent, adsorbed] {PCV10} were administered in a 2+1 regimen (ie, 2 doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5 MoA] and 1 final dose in the second year of life [12 to 18 MoA]); and the measles, mumps, rubella (MMR) vaccine was administered at 12 to 18 MoA.
  Interventions: Biological: MenACYW conjugate vaccine; Biological: DTaP-IPV-HB-Hib vaccine; Biological: Pneumococcal vaccine (10-valent); Biological: MMR vaccine
- Group 2: Nimenrix (Active Comparator): Participants received 3 doses of Nimenrix® 0.5 mL as an IM injection at dose 1: 2 MoA, dose 2: 4 MoA, and dose 3: 12 to 18 MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (DTaP-IPV-HB-Hib), the PCV10 were administered in a 2+1 regimen (ie, 2 doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5 MoA] and 1 final dose in the second year of life [12 to 18 MoA]); and the MMR vaccine was administered at 12 to 18 MoA.
  Interventions: Biological: Meningococcal group A, C, W-135, and Y conjugate vaccine; Biological: DTaP-IPV-HB-Hib vaccine; Biological: Pneumococcal vaccine (10-valent); Biological: MMR vaccine
- Group 3: MenACYW (Experimental): Participants received 3 doses of MenACYW conjugate vaccine 0.5 mL as an IM injection at dose 1: 2 MoA, dose 2: 4 MoA, and dose 3: 12 to 18 MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (DTaP-IPV-HB-Hib), the pneumococcal conjugate vaccine (13-valent, adsorbed) [PCV13] were administered in a 2+1 regimen (ie, 2 doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5 MoA] and 1 final dose in the second year of life [12 to 18 MoA]); and the MMR vaccine was administered at 12 to 18 MoA.
  Interventions: Biological: MenACYW conjugate vaccine; Biological: DTaP-IPV-HB-Hib vaccine; Biological: Pneumococcal vaccine (13-valent); Biological: MMR vaccine
- Group 4: MenACYW (Experimental): Participants received 4 doses of MenACYW conjugate vaccine 0.5 mL as an IM injection at dose 1: 2 MoA, dose 2: 4 MoA, and dose 3: 6 MoA and dose 4: 12 to 18 MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (DTaP-IPV-HB-Hib), the PCV13 were administered in a 2+1 regimen (concomitantly with the first and second doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5 MoA] and the toddler dose of MenACYW conjugate vaccine [12 to 18 MoA]); and the MMR vaccine was administered at 12 to 18 MoA. The third dose of MenACYW conjugate vaccine was administered alone, without any other routine pediatric vaccines.
  Interventions: Biological: MenACYW conjugate vaccine; Biological: DTaP-IPV-HB-Hib vaccine; Biological: Pneumococcal vaccine (13-valent); Biological: MMR vaccine

INTERVENTIONS:
Biological: MenACYW conjugate vaccine — Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine, 0.5 mL, intramuscular
  Other Names: MenQuadfi®
  Arms: Group 1: MenACYW; Group 3: MenACYW; Group 4: MenACYW
Biological: Meningococcal group A, C, W-135, and Y conjugate vaccine — Meningococcal group A, C, W-135, and Y conjugate vaccine, 0.5 mL, intramuscular
  Other Names: Nimenrix®
  Arms: Group 2: Nimenrix
Biological: DTaP-IPV-HB-Hib vaccine — Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type b vaccine
  Other Names: Hexyon®/Hexacima®
Biological: Pneumococcal vaccine (13-valent) — Pneumococcal polysaccharide conjugate vaccine (13-valent, adsorbed)
  Other Names: Prevenar 13®
  Arms: Group 3: MenACYW; Group 4: MenACYW
Biological: Pneumococcal vaccine (10-valent) — Pneumococcal polysaccharide conjugate vaccine (10-valent, adsorbed)
  Other Names: Synflorix®
  Arms: Group 1: MenACYW; Group 2: Nimenrix
Biological: MMR vaccine — Measles, mumps, and rubella vaccine
  Other Names: M-M-RVAXPRO®

SUMMARY:
Primary objective:

This study aimed to demonstrate the non-inferiority of the antibody response against meningococcal serogroups A, C, Y, and W following the administration of a 3-dose series of MenACYW conjugate vaccine compared to a 3-dose series of a licensed meningococcal vaccine when each vaccine was given concomitantly with routine pediatric vaccines (10-valent pneumococcal vaccine and diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type b [DTaP-IPV-HB-Hib vaccine]) to infants and toddlers 6 weeks to 18 months old

Secondary objectives:

This study aimed to demonstrate the non-inferiority of the antibody (Ab) response against meningococcal serogroups A, C, Y, and W following the administration of 2 doses in infancy of MenACYW conjugate vaccine compared to 2 doses of a licensed meningococcal vaccine when each vaccine was given concomitantly with routine pediatric vaccines (10-valent pneumococcal vaccine and DTaP-IPV-HB-Hib vaccine) to infants and toddlers 6 weeks to 18 months old.

- This study aimed to describe the Ab responses against meningococcal groups A, C, Y, and W and the antigens of the routine pediatric vaccines administered in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 42 to ≤ 89 days on the day of the first study visit
* Healthy infants as determined by medical history, physical examination and judgment of the Investigator
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative
* Subject and parent/legally acceptable representative were able to attend all scheduled visits and to comply with all study procedures
* Covered by health insurance according to local regulations

Exclusion Criteria:

* Participated at the time of study enrollment (or in the 4 weeks preceding the first study vaccination) or planned participation during the study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Received any vaccine in the 4 weeks preceding the first study vaccination or planned receipt of any vaccine in the 4 weeks before and/or following any study vaccination except for influenza vaccination and rotavirus vaccination, which may be received at a gap of at least 2 weeks before or 2 weeks after any study vaccines. This exception included monovalent pandemic influenza vaccines and multivalent influenza vaccines. This exclusion criterion did not apply to subjects in Finland, Sweden or Poland who planned to receive the licensed rotavirus vaccine concomitantly with study vaccines at study vaccination visits V1 and V2.
* Received or planned to receipt during the study period vaccination against meningococcal disease with either the study vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B serogroup-containing vaccine)
* Previous vaccination against diphtheria, tetanus, pertussis, Haemophilus influenzae type B (Hib), poliovirus, Streptococcus pneumoniae, measles, mumps, or rubella. Previous vaccination against hepatitis B when administered to risk groups, as per local recommendation.
* Received immune globulins, blood or blood-derived products since birth
* Known or suspected congenital or acquired immunodeficiency; or received immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) since birth
* Family history of congenital or hereditary immunodeficiency, unless the immune competence of the potential vaccine recipient is demonstrated
* Individuals that had blood dyscrasias, leukemia, lymphoma of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems
* Individuals that had active tuberculosis
* History of Neisseria meningitidis infection, confirmed either clinically, serologically, or microbiologically
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, measles, mumps, rubella, and of Haemophilus influenzae type b, and / or Streptococcus pneumoniae infection or disease
* Individuals that were at high risk for meningococcal infection during the study (specifically, but not limited to, subjects that had persistent complement deficiency, with anatomic or functional asplenia, or subjects traveling to countries with high endemic or epidemic disease)
* Individuals that had underlying conditions predisposing them to invasive pneumococcal disease (specifically, but not limited to, subjects with sickle cell disease or human immunodeficiency virus [HIV] infection)
* History of any neurologic disorders, including seizures and progressive neurologic disorders
* History of Guillain-Barré syndrome
* Known systemic hypersensitivity to any of the vaccine components, or history of a severe allergic reaction (e.g., anaphylaxis) to the vaccine(s) used in the study or to a vaccine containing any of the same substances including neomycin, streptomycin, polymyxin B, glutaraldehyde, formaldehyde, and gelatin
* Reported of thrombocytopenia, contraindicating intramuscular vaccination in the investigator's opinion
* Bleeding disorder, or received of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the investigator's opinion
* Chronic illness (including, but not limited to, cardiac disorders, congenital heart disease, chronic lung disease, renal disorders, auto-immune disorders, diabetes, psychomotor diseases, and known congenital or genetic diseases) that, in the opinion of the investigator, were at a stage where it could interfere with study conduct or completion
* Any condition which, in the opinion of the investigator, could interfere with the evaluation of the study objectives, including planned to leave the area of the study site before the end of the study
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective subject could not be included in the study until the condition was resolved or the febrile event was subsided.
* Received oral or injectable antibiotic therapy within 72 hours prior to the first blood draw Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study
* Infants born preterm (by less than 37 weeks of gestation) required specific immunization schedule for routine childhood vaccines and/or specific care at the time of vaccination, as per national recommendations

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1660 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (33):
- Czechia (9):
  - Investigational Site Number : 2031006, Chlumec nad Cidlinou
  - Investigational Site Number : 2031013, Domažlice
  - Investigational Site Number : 2031010, Jindřichův Hradec
  - Investigational Site Number : 2031012, Jindřichův Hradec
  - Investigational Site Number : 2031003, Ostrava
  - Investigational Site Number : 2031008, Ostrava-hrabuvka
  - Investigational Site Number : 2031009, Pardubice
  - Investigational Site Number : 2031005, Pardubice
  - Investigational Site Number : 2031007, Smiřice
- Finland (10):
  - Investigational Site Number : 2462007, Espoo
  - Investigational Site Number : 2462003, Helsinki
  - Investigational Site Number : 2462004, Helsinki
  - Investigational Site Number : 2462001, Jarvenpaa
  - Investigational Site Number : 2462006, Kokkola
  - Investigational Site Number : 2462005, Oulu
  - Investigational Site Number : 2462002, Pori
  - Investigational Site Number : 2462009, Seinäjoki
  - Investigational Site Number : 2462010, Tampere
  - Investigational Site Number : 2462008, Turku
- Investigational Site Number : 3803002, Milan, Italy
- Poland (4):
  - Investigational Site Number : 6167002, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6167004, Trzebnica, Lower Silesian Voivodeship
  - Investigational Site Number : 6167003, Siemianowice Śląskie
  - Investigational Site Number : 6167006, Torun
- Romania (4):
  - Investigational Site Number : 6424003, Brasov
  - Investigational Site Number : 6424001, Bucaresti
  - Investigational Site Number : 6424006, Caracal
  - Investigational Site Number : 6424002, Călăraşi
- Spain (4):
  - Investigational Site Number : 7245003, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7245002, Madrid
  - Investigational Site Number : 7245001, Santiago de Compostela
  - Investigational Site Number : 7245006, Seville
- Investigational Site Number : 7526001, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Martinon-Torres F, Virta MM, Koski S, de la Cueva IS, Szymanski HT, Bosis S, Draganescu AC, Silfverdal SA, Zambrano B, Dhingra MS, B'Chir S, Syrkina O, Lyabis O, Vasquez GA, Rehm C; MET58 Study Group. Immunogenicity and Safety of a Quadrivalent Meningococcal Conjugate Vaccine (MenACYW-TT) Administered with Routine Pediatric Vaccines: A European Randomized Controlled Trial. Infect Dis Ther. 2025 Aug;14(8):1843-1865. doi: 10.1007/s40121-025-01190-7. Epub 2025 Jul 15. PMID 40665158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 33 investigational sites in 7 countries between 14 December 2018 to 24 May 2023.
Pre-assignment Details: A total of 1660 participants were enrolled in this study.
Period: Overall Study
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Started | 714 | 726 | 112 | 108
Safety Analysis Set (SafAS) | 696 | 706 | 112 | 108
Completed | 681 | 691 | 106 | 104
Not Completed | 33 | 35 | 6 | 4
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Protocol deviation | 5 | 7 | 3 | 0
Not completed — Withdrawal by Parent/Guardian | 24 | 24 | 2 | 4
Not completed — Lost to Follow-up | 3 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants included study participants for whom an injection group had been allocated.
Groups:
- Group 1: MenACYW: Participants received 3 doses of MenACYW conjugate vaccine 0.5 mL as an IM injection at dose 1: 2 MoA, dose 2: 4 MoA, and dose 3: 12 to 18 MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (DTaP-IPV-HB-Hib), the PCV10 were administered in a 2+1 regimen (ie, 2 doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5 MoA] and 1 final dose in the second year of life [12 to 18 MoA]); and the MMR vaccine was administered at 12 to 18 MoA.
- Group 3: MenACYW: Participants received 3 doses of MenACYW conjugate vaccine 0.5 mL as an IM injection at dose 1: 2 MoA, dose 2: 4 MoA, and dose 3: 12 to 18 MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (DTaP-IPV-HB-Hib), the PCV13 were administered in a 2+1 regimen (ie, 2 doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5 MoA] and 1 final dose in the second year of life [12 to 18 MoA]); and the MMR vaccine was administered at 12 to 18 MoA.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW | Total
Number analyzed (Participants) | 714 | 726 | 112 | 108 | 1660
Age, Continuous [Mean (Standard Deviation); unit: Days] | 72.6 (12.2) | 72.4 (12.1) | 62.5 (7.12) | 63.3 (7.93) | 71.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 355 | 378 | 45 | 58 | 836
  Male | 359 | 348 | 67 | 50 | 824
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 4 | 2 | 9
  Black or African American | 0 | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  White | 693 | 699 | 106 | 101 | 1599
  Not Reported | 13 | 16 | 0 | 1 | 30
  Unknown | 2 | 3 | 0 | 0 | 5
  Multiple origin | 4 | 6 | 0 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Groups 1 and 2: Geometric Mean Titers (GMTs) Against Meningococcal Serogroups A, C, W, and Y
Description: Functional meningococcal antibody activity against serogroups A, C, W, and Y were measured in a serum bactericidal assay utilizing the serum bactericidal assay using human complement (hSBA).
Time Frame: At 30 days post Dose 3 [12 to 18 months of age (MoA)]
Population: Per-Protocol Analysis Set 2 (PPAS2) was a subset of Full Analysis Set 2 (FAS2). The FAS2 included the subset of randomized participants who received at least 1 dose of the study vaccine at booster vaccination and had a valid post-booster vaccination blood sample result. Only participants with data collected for each specific serogroup are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix
Number analyzed (Participants) | 554 | 579
Titer
  Serogroup A: number analyzed (Participants) | 543 | 567
  Serogroup A | 131 [113 to 151] | 189 [165 to 218]
  Serogroup C: number analyzed (Participants) | 550 | 578
  Serogroup C | 565 [505 to 632] | 120 [106 to 135]
  Serogroup W: number analyzed (Participants) | 547 | 575
  Serogroup W | 423 [382 to 468] | 275 [247 to 305]
  Serogroup Y | 285 [260 to 313] | 160 [145 to 177]
Statistical Analysis 1: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup A; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) was >1/1.5 for all 4 serogroups; GMT ratio = 0.690, 95% CI 2-sided [0.565 to 0.842] — 95% CI of the GMT ratio was calculated using a normal approximation of log-transformed titers
Statistical Analysis 2: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup C; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >1/1.5 for all 4 serogroups; GMT ratio = 4.73, 95% CI 2-sided [4.00 to 5.58] — 95% CI of the GMT ratio was calculated using a normal approximation of log-transformed titers
Statistical Analysis 3: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup W; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >1/1.5 for all 4 serogroups; Slope = 1.54, 95% CI 2-sided [1.33 to 1.78] — 95% CI of the GMT ratio was calculated using a normal approximation of log-transformed titers
Statistical Analysis 4: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup Y; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >1/1.5 for all 4 serogroups; GMT ratio = 1.78, 95% CI 2-sided [1.55 to 2.04] — 95% CI of the GMT ratio was calculated using a normal approximation of log-transformed titers

2. Secondary Outcome: Groups 1 and 2: Percentage of Participants Who Achieved Antibody Titers >=1:8 Against Meningococcal Serogroups A, C, W, and Y
Description: Functional meningococcal antibody activity against serogroups A, C, W, and Y were measured in a serum bactericidal assay utilizing the hSBA. Percentages are rounded off to the tenth decimal place.
Time Frame: At 30 days post Dose 2 (4 MoA)
Population: PPAS1 was a subset of FAS1. The FAS1 included the subset of randomized participants who received at least 1 dose of the study vaccine in the primary series and had a valid post-primary series vaccination blood sample result. Only participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix
Number analyzed (Participants) | 518 | 523
Percentage of participants
  Serogroup A: number analyzed (Participants) | 508 | 508
  Serogroup A | 63.6 [59.2 to 67.8] | 75.8 [71.8 to 79.5]
  Serogroup C: number analyzed (Participants) | 513 | 521
  Serogroup C | 98.8 [97.5 to 99.6] | 91.9 [89.3 to 94.1]
  Serogroup W | 96.5 [94.6 to 97.9] | 94.5 [92.1 to 96.3]
  Serogroup Y: number analyzed (Participants) | 516 | 523
  Serogroup Y | 96.5 [94.5 to 97.9] | 93.5 [91.0 to 95.5]
Statistical Analysis 1: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup A; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for all 4 serogroups; Difference in percentage of participants = -12.20, 95% CI 2-sided [-17.74 to -6.56] — 95% CI of the difference was calculated from the Wilson score method without continuity correction
Statistical Analysis 2: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup C; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for all 4 serogroups; Difference in percentage of participants = 6.89, 95% CI 2-sided [4.44 to 9.62] — 95% CI of the difference was calculated from the Wilson score method without continuity correction
Statistical Analysis 3: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup W; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for all 4 serogroups; Difference in percentage of participants = 2.07, 95% CI 2-sided [-0.49 to 4.70] — 95% CI of the difference was calculated from the Wilson score method without continuity correction
Statistical Analysis 4: Comparison: Group 1: MenACYW vs Group 2: Nimenrix; Statistical analysis for Serogroup Y; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for all 4 serogroups; Difference in percentage of participants = 3.01, 95% CI 2-sided [0.34 to 5.77] — 95% CI of the difference was calculated from the Wilson score method without continuity correction

3. Secondary Outcome: Groups 3 and 4: Geometric Mean Titers (GMTs) Against Meningococcal Serogroups A, C, W, and Y
Description: Functional meningococcal antibody activity against serogroups A, C, W, and Y were measured in a serum bactericidal assay utilizing the hSBA.
Time Frame: Group 3: Day 0 before Dose 1 (2 MoA) and Dose 3 (12 to 18 MoA) and Day 30 Post Dose 2 (4 MoA) and Dose 3 (12 to 18 MoA); Group 4: Day 0 before Dose 1 (2 MoA) and Dose 4 (12 to 18 MoA) and Day 30 Post Dose 3 (6 MoA) and Dose 4 (12 to 18 MoA)
Population: PPAS1 was a subset of FAS1. FAS1: subset of randomized participants who received at least 1 dose of study vaccine in primary series and had valid post-primary series vaccination blood sample result. PPAS2 was a subset of FAS2. FAS2: subset of randomized participants who received at least 1 dose of study vaccine at booster vaccination and had valid post-booster vaccination blood sample result. Only participants with data collected for each specific serogroup at specified timepoints are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 96 | 90
Titer
  PPAS1: Serogroup A: Day 0 before dose 1: number analyzed (Participants) | 94 | 89
  PPAS1: Serogroup A: Day 0 before dose 1 | 3.00 [2.58 to 3.49] | 2.86 [2.49 to 3.28]
  PPAS1: Serogroup A: Day 30 post dose 2: number analyzed (Participants) | 91 | 0
  PPAS1: Serogroup A: Day 30 post dose 2 | 14.8 [10.6 to 20.8] |
  PPAS1: Serogroup A: Day 30 post dose 3: number analyzed (Participants) | 0 | 88
  PPAS1: Serogroup A: Day 30 post dose 3 |  | 23.0 [17.1 to 30.9]
  PPAS1: Serogroup C: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup C: Day 0 before dose 1 | 3.91 [3.16 to 4.84] | 3.88 [3.25 to 4.62]
  PPAS1: Serogroup C: Day 30 post dose 2: number analyzed (Participants) | 95 | 0
  PPAS1: Serogroup C: Day 30 post dose 2 | 309 [235 to 407] |
  PPAS1: Serogroup C: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup C: Day 30 post dose 3 |  | 481 [376 to 616]
  PPAS1: Serogroup W: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup W: Day 0 before dose 1 | 2.67 [2.40 to 2.96] | 3.08 [2.63 to 3.60]
  PPAS1: Serogroup W: Day 30 post dose 2: number analyzed (Participants) | 96 | 0
  PPAS1: Serogroup W: Day 30 post dose 2 | 102 [79.7 to 131] |
  PPAS1: Serogroup W: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup W: Day 30 post dose 3 |  | 196 [156 to 245]
  PPAS1: Serogroup Y: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup Y: Day 0 before dose 1 | 2.85 [2.45 to 3.32] | 2.76 [2.36 to 3.23]
  PPAS1: Serogroup Y: Day 30 post dose 2: number analyzed (Participants) | 96 | 0
  PPAS1: Serogroup Y: Day 30 post dose 2 | 73.4 [57.7 to 93.5] |
  PPAS1: Serogroup Y: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup Y: Day 30 post dose 3 |  | 150 [116 to 195]
  PPAS2: Serogroup A: Day 0 before dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup A: Day 0 before dose 3 | 5.18 [4.22 to 6.37] |
  PPAS2: Serogroup A: Day 30 post dose 3: number analyzed (Participants) | 92 | 0
  PPAS2: Serogroup A: Day 30 post dose 3 | 104 [67.9 to 161] |
  PPAS2: Serogroup A: Day 0 before dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup A: Day 0 before dose 4 |  | 8.13 [6.33 to 10.4]
  PPAS2: Serogroup A: Day 30 post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup A: Day 30 post dose 4 |  | 62.0 [39.9 to 96.4]
  PPAS2: Serogroup C: Day 0 before dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup C: Day 0 before dose 3 | 26.2 [18.7 to 36.8] |
  PPAS2: Serogroup C: Day 30 post dose 3: number analyzed (Participants) | 93 | 0
  PPAS2: Serogroup C: Day 30 post dose 3 | 819 [622 to 1078] |
  PPAS2: Serogroup C: Day 0 before dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup C: Day 0 before dose 4 |  | 56.9 [42.4 to 76.4]
  PPAS2: Serogroup C: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup C: Day 30 post dose 4 |  | 791 [608 to 1029]
  PPAS2: Serogroup W: Day 0 before dose 3: number analyzed (Participants) | 93 | 0
  PPAS2: Serogroup W: Day 0 before dose 3 | 39.1 [29.6 to 51.8] |
  PPAS2: Serogroup W: Day 30 post dose 3: number analyzed (Participants) | 87 | 0
  PPAS2: Serogroup W: Day 30 post dose 3 | 1049 [782 to 1406] |
  PPAS2: Serogroup W: Day 0 before dose 4: number analyzed (Participants) | 0 | 90
  PPAS2: Serogroup W: Day 0 before dose 4 |  | 92.6 [74.3 to 115]
  PPAS2: Serogroup W: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup W: Day 30 post dose 4 |  | 1024 [806 to 1301]
  PPAS2: Serogroup Y: Day 0 before dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup Y: Day 0 before dose 3 | 33.0 [25.0 to 43.5] |
  PPAS2: Serogroup Y: Day 30 post dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup Y: Day 30 post dose 3 | 589 [470 to 737] |
  PPAS2: Serogroup Y: Day 0 before dose 4: number analyzed (Participants) | 0 | 90
  PPAS2: Serogroup Y: Day 0 before dose 4 |  | 85.8 [68.2 to 108]
  PPAS2: Serogroup Y: Day 30 post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup Y: Day 30 post dose 4 |  | 632 [512 to 780]

4. Secondary Outcome: Groups 1 and 2: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Antibody Titers >=1:4 and >=1:8
Description: as for outcome 2
Time Frame: Day 0 Before Dose 1 (2 MoA) and Day 30 Post Dose 2 (4 MoA); Day 0 Before Dose 3 (12 to 18 MoA) and Day 30 Post Dose 3 (12 to 18 MoA)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 1: MenACYW: Participants received 3 doses of MenACYW conjugate vaccine 0.5 mL as an IM injection at dose 1: 2 MoA, dose 2: 4 MoA, and dose 3: 12 to 18MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (DTaP-IPV-HB-Hib), thePCV10 were administered in a 2+1 regimen (ie, 2 doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5 MoA] and 1 final dose in the second year of life [12 to 18 MoA]); and the MMR vaccine was administeredat 12 to 18 MoA.
- Group 2: Nimenrix: Participants received 3 doses of Nimenrix® 0.5 mL as an IM injection at dose 1: 2 MoA, dose 2: 4 MoA, and dose 3: 12 to 18 MoA along with routine pediatric vaccines. The routine pediatric vaccines: hexavalent vaccine (DTaP-IPV-HB-Hib), the PCV10 were administered in a 2+1 regimen (ie, 2 doses in infancy [first between 6 and 12 weeks of age and second between 4 to 5MoA] and 1 final dose in the second year of life [12 to 18 MoA]); and the MMR vaccine was administered at 12 to 18 MoA.
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix
Number analyzed (Participants) | 554 | 579
Percentage of participants
  PPAS1: Serogroup A: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 521 | 519
  PPAS1: Serogroup A: >=1:4: Day 0 before dose 1 | 31.1 [27.1 to 35.3] | 28.3 [24.5 to 32.4]
  PPAS1: Serogroup A: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 521 | 519
  PPAS1: Serogroup A: >=1:8: Day 0 before dose 1 | 5.6 [3.8 to 7.9] | 6.4 [4.4 to 8.8]
  PPAS1: Serogroup A: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 508 | 508
  PPAS1: Serogroup A: >=1:4: Day 30 post dose 2 | 77.2 [73.3 to 80.7] | 88.0 [84.8 to 90.7]
  PPAS1: Serogroup A: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 508 | 508
  PPAS1: Serogroup A: >=1:8: Day 30 post dose 2 | 63.6 [59.2 to 67.8] | 75.8 [71.8 to 79.5]
  PPAS1: Serogroup C: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 517 | 517
  PPAS1: Serogroup C: >=1:4: Day 0 before dose 1 | 14.3 [11.4 to 17.6] | 14.9 [11.9 to 18.3]
  PPAS1: Serogroup C: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 517 | 517
  PPAS1: Serogroup C: >=1:8: Day 0 before dose 1 | 5.2 [3.5 to 7.5] | 5.2 [3.5 to 7.5]
  PPAS1: Serogroup C: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 513 | 521
  PPAS1: Serogroup C: >=1:4: Day 30 post dose 2 | 99.0 [97.7 to 99.7] | 96.4 [94.4 to 97.8]
  PPAS1: Serogroup C: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 513 | 521
  PPAS1: Serogroup C: >=1:8: Day 30 post dose 2 | 98.8 [97.5 to 99.6] | 91.9 [89.3 to 94.1]
  PPAS1: Serogroup W: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 520 | 520
  PPAS1: Serogroup W: >=1:4: Day 0 before dose 1 | 11.7 [9.1 to 14.8] | 11.0 [8.4 to 14.0]
  PPAS1: Serogroup W: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 520 | 520
  PPAS1: Serogroup W: >=1:8: Day 0 before dose 1 | 3.7 [2.2 to 5.6] | 3.5 [2.1 to 5.4]
  PPAS1: Serogroup W: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 518 | 523
  PPAS1: Serogroup W: >=1:4: Day 30 post dose 2 | 98.6 [97.2 to 99.5] | 98.3 [96.8 to 99.2]
  PPAS1: Serogroup W: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 518 | 523
  PPAS1: Serogroup W: >=1:8: Day 30 post dose 2 | 96.5 [94.6 to 97.9] | 94.5 [92.1 to 96.3]
  PPAS1: Serogroup Y: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 519 | 518
  PPAS1: Serogroup Y: >=1:4: Day 0 before dose 1 | 10.0 [7.6 to 12.9] | 9.8 [7.4 to 12.7]
  PPAS1: Serogroup Y: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 519 | 518
  PPAS1: Serogroup Y: >=1:8: Day 0 before dose 1 | 6.4 [4.4 to 8.8] | 5.6 [3.8 to 7.9]
  PPAS1: Serogroup Y: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 516 | 523
  PPAS1: Serogroup Y: >=1:4: Day 30 post dose 2 | 98.3 [96.7 to 99.2] | 97.3 [95.5 to 98.5]
  PPAS1: Serogroup Y: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 516 | 523
  PPAS1: Serogroup Y: >=1:8: Day 30 post dose 2 | 96.5 [94.5 to 97.9] | 93.5 [91.0 to 95.5]
  PPAS2: Serogroup A: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 540 | 567
  PPAS2: Serogroup A: >=1:4: Day 0 before dose 3 | 69.1 [65.0 to 73.0] | 73.7 [69.9 to 77.3]
  PPAS2: Serogroup A: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 540 | 567
  PPAS2: Serogroup A: >=1:8: Day 0 before dose 3 | 33.7 [29.7 to 37.9] | 46.2 [42.0 to 50.4]
  PPAS2: Serogroup A: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 543 | 567
  PPAS2: Serogroup A: >=1:4: Day 30 post dose 3 | 98.2 [96.6 to 99.1] | 98.1 [96.6 to 99.0]
  PPAS2: Serogroup A: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 543 | 567
  PPAS2: Serogroup A: >=1:8: Day 30 post dose 3 | 94.7 [92.4 to 96.4] | 96.5 [94.6 to 97.8]
  PPAS2: Serogroup C: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 545 | 572
  PPAS2: Serogroup C: >=1:4: Day 0 before dose 3 | 92.5 [89.9 to 94.5] | 62.1 [57.9 to 66.1]
  PPAS2: Serogroup C: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 545 | 572
  PPAS2: Serogroup C: >=1:8: Day 0 before dose 3 | 88.1 [85.1 to 90.7] | 41.6 [37.5 to 45.8]
  PPAS2: Serogroup C: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 550 | 578
  PPAS2: Serogroup C: >=1:4: Day 30 post dose 3 | 99.8 [99.0 to 100] | 98.1 [96.6 to 99.0]
  PPAS2: Serogroup C: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 550 | 578
  PPAS2: Serogroup C: >=1:8: Day 30 post dose 3 | 99.6 [98.7 to 100] | 95.5 [93.5 to 97.0]
  PPAS2: Serogroup W: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 541 | 567
  PPAS2: Serogroup W: >=1:4: Day 0 before dose 3 | 96.7 [94.8 to 98.0] | 91.2 [88.5 to 93.4]
  PPAS2: Serogroup W: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 541 | 567
  PPAS2: Serogroup W: >=1:8: Day 0 before dose 3 | 89.1 [86.2 to 91.6] | 77.6 [73.9 to 81.0]
  PPAS2: Serogroup W: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 547 | 575
  PPAS2: Serogroup W: >=1:4: Day 30 post dose 3 | 100 [99.3 to 100] | 100 [99.4 to 100]
  PPAS2: Serogroup W: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 547 | 575
  PPAS2: Serogroup W: >=1:8: Day 30 post dose 3 | 99.8 [99.0 to 100] | 99.5 [98.5 to 99.9]
  PPAS2: Serogroup Y: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 545 | 572
  PPAS2: Serogroup Y: >=1:4: Day 0 before dose 3 | 95.8 [93.7 to 97.3] | 85.7 [82.5 to 88.4]
  PPAS2: Serogroup Y: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 545 | 572
  PPAS2: Serogroup Y: >=1:8: Day 0 before dose 3 | 87.9 [84.9 to 90.5] | 69.6 [65.6 to 73.3]
  PPAS2: Serogroup Y: >=1:4: Day 30 post dose 3 | 100 [99.3 to 100] | 100 [99.4 to 100]
  PPAS2: Serogroup Y: >=1:8: Day 30 post dose 3 | 100 [99.3 to 100] | 99.8 [99.0 to 100]

5. Secondary Outcome: Groups 3 and 4: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Antibody Titers >=1:4 and >=1:8
Description: as for outcome 2
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 96 | 90
Percentage of participants
  PPAS1: Serogroup A: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 94 | 89
  PPAS1: Serogroup A: >=1:4: Day 0 before dose 1 | 33.0 [23.6 to 43.4] | 32.6 [23.0 to 43.3]
  PPAS1: Serogroup A: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 94 | 89
  PPAS1: Serogroup A: >=1:8: Day 0 before dose 1 | 14.9 [8.4 to 23.7] | 11.2 [5.5 to 19.7]
  PPAS1: Serogroup A: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 91 | 0
  PPAS1: Serogroup A: >=1:4: Day 30 post dose 2 | 79.1 [69.3 to 86.9] |
  PPAS1: Serogroup A: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 91 | 0
  PPAS1: Serogroup A: >=1:8: Day 30 post dose 2 | 63.7 [53.0 to 73.6] |
  PPAS1: Serogroup A: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 0 | 88
  PPAS1: Serogroup A: >=1:4: Day 30 post dose 3 |  | 92.0 [84.3 to 96.7]
  PPAS1: Serogroup A: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 0 | 88
  PPAS1: Serogroup A: >=1:8: Day 30 post dose 3 |  | 81.8 [72.2 to 89.2]
  PPAS1: Serogroup C: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup C: >=1:4: Day 0 before dose 1 | 43.6 [33.4 to 54.2] | 48.9 [38.2 to 59.7]
  PPAS1: Serogroup C: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup C: >=1:8: Day 0 before dose 1 | 26.6 [18.0 to 36.7] | 32.2 [22.8 to 42.9]
  PPAS1: Serogroup C: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 95 | 0
  PPAS1: Serogroup C: >=1:4: Day 30 post dose 2 | 98.9 [94.3 to 100] |
  PPAS1: Serogroup C: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 95 | 0
  PPAS1: Serogroup C: >=1:8: Day 30 post dose 2 | 98.9 [94.3 to 100] |
  PPAS1: Serogroup C: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup C: >=1:4: Day 30 post dose 3 |  | 98.9 [94.0 to 100]
  PPAS1: Serogroup C: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup C: >=1:8: Day 30 post dose 3 |  | 98.9 [94.0 to 100]
  PPAS1: Serogroup W: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup W: >=1:4: Day 0 before dose 1 | 28.7 [19.9 to 39.0] | 35.6 [25.7 to 46.3]
  PPAS1: Serogroup W: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup W: >=1:8: Day 0 before dose 1 | 10.6 [5.2 to 18.7] | 16.7 [9.6 to 26.0]
  PPAS1: Serogroup W: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 96 | 0
  PPAS1: Serogroup W: >=1:4: Day 30 post dose 2 | 99.0 [94.3 to 100] |
  PPAS1: Serogroup W: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 96 | 0
  PPAS1: Serogroup W: >=1:8: Day 30 post dose 2 | 96.9 [91.1 to 99.4] |
  PPAS1: Serogroup W: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup W: >=1:4: Day 30 post dose 3 |  | 98.9 [94.0 to 100]
  PPAS1: Serogroup W: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup W: >=1:8: Day 30 post dose 3 |  | 98.9 [94.0 to 100]
  PPAS1: Serogroup Y: >=1:4: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup Y: >=1:4: Day 0 before dose 1 | 26.6 [18.0 to 36.7] | 22.2 [14.1 to 32.2]
  PPAS1: Serogroup Y: >=1:8: Day 0 before dose 1: number analyzed (Participants) | 94 | 90
  PPAS1: Serogroup Y: >=1:8: Day 0 before dose 1 | 12.8 [6.8 to 21.2] | 12.2 [6.3 to 20.8]
  PPAS1: Serogroup Y: >=1:4: Day 30 post dose 2: number analyzed (Participants) | 96 | 0
  PPAS1: Serogroup Y: >=1:4: Day 30 post dose 2 | 99.0 [94.3 to 100] |
  PPAS1: Serogroup Y: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 96 | 0
  PPAS1: Serogroup Y: >=1:8: Day 30 post dose 2 | 95.8 [89.7 to 98.9] |
  PPAS1: Serogroup Y: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup Y: >=1:4: Day 30 post dose 3 |  | 98.9 [94.0 to 100]
  PPAS1: Serogroup Y: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup Y: >=1:8: Day 30 post dose 3 |  | 98.9 [94.0 to 100]
  PPAS2: Serogroup A: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup A: >=1:4: Day 0 before dose 3 | 65.9 [55.3 to 75.5] |
  PPAS2: Serogroup A: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup A: >=1:8: Day 0 before dose 3 | 37.4 [27.4 to 48.1] |
  PPAS2: Serogroup A: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 92 | 0
  PPAS2: Serogroup A: >=1:4: Day 30 post dose 3 | 92.4 [84.9 to 96.9] |
  PPAS2: Serogroup A: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 92 | 0
  PPAS2: Serogroup A: >=1:8: Day 30 post dose 3 | 89.1 [80.9 to 94.7] |
  PPAS2: Serogroup A: >=1:4: Day 0 before dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup A: >=1:4: Day 0 before dose 4 |  | 80.9 [71.2 to 88.5]
  PPAS2: Serogroup A: >=1:8: Day 0 before dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup A: >=1:8: Day 0 before dose 4 |  | 52.8 [41.9 to 63.5]
  PPAS2: Serogroup A: >=1:4: Day 30 post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup A: >=1:4: Day 30 post dose 4 |  | 82.0 [72.5 to 89.4]
  PPAS2: Serogroup A: >=1:8: Day 30 post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup A: >=1:8: Day 30 post dose 4 |  | 82.0 [72.5 to 89.4]
  PPAS2: Serogroup C: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup C: >=1:4: Day 0 before dose 3 | 87.2 [78.8 to 93.2] |
  PPAS2: Serogroup C: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup C: >=1:8: Day 0 before dose 3 | 79.8 [70.2 to 87.4] |
  PPAS2: Serogroup C: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 93 | 0
  PPAS2: Serogroup C: >=1:4: Day 30 post dose 3 | 100 [96.1 to 100] |
  PPAS2: Serogroup C: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 93 | 0
  PPAS2: Serogroup C: >=1:8: Day 30 post dose 3 | 100 [96.1 to 100] |
  PPAS2: Serogroup C: >=1:4: Day 0 before dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup C: >=1:4: Day 0 before dose 4 |  | 97.8 [92.1 to 99.7]
  PPAS2: Serogroup C: >=1:8: Day 0 before dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup C: >=1:8: Day 0 before dose 4 |  | 92.1 [84.5 to 96.8]
  PPAS2: Serogroup C: >=1:4: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup C: >=1:4: Day 30 post dose 4 |  | 100 [95.8 to 100]
  PPAS2: Serogroup C: >=1:8: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup C: >=1:8: Day 30 post dose 4 |  | 100 [95.8 to 100]
  PPAS2: Serogroup W: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 93 | 0
  PPAS2: Serogroup W: >=1:4: Day 0 before dose 3 | 96.8 [90.9 to 99.3] |
  PPAS2: Serogroup W: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 93 | 0
  PPAS2: Serogroup W: >=1:8: Day 0 before dose 3 | 92.5 [85.1 to 96.9] |
  PPAS2: Serogroup W: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 87 | 0
  PPAS2: Serogroup W: >=1:4: Day 30 post dose 3 | 100 [95.8 to 100] |
  PPAS2: Serogroup W: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 87 | 0
  PPAS2: Serogroup W: >=1:8: Day 30 post dose 3 | 100 [95.8 to 100] |
  PPAS2: Serogroup W: >=1:4: Day 0 before dose 4: number analyzed (Participants) | 0 | 90
  PPAS2: Serogroup W: >=1:4: Day 0 before dose 4 |  | 100 [96.0 to 100]
  PPAS2: Serogroup W: >=1:8: Day 0 before dose 4: number analyzed (Participants) | 0 | 90
  PPAS2: Serogroup W: >=1:8: Day 0 before dose 4 |  | 100 [96.0 to 100]
  PPAS2: Serogroup W: >=1:4: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup W: >=1:4: Day 30 post dose 4 |  | 100 [95.8 to 100]
  PPAS2: Serogroup W: >=1:8: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup W: >=1:8: Day 30 post dose 4 |  | 100 [95.8 to 100]
  PPAS2: Serogroup Y: >=1:4: Day 0 before dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup Y: >=1:4: Day 0 before dose 3 | 94.7 [88.0 to 98.3] |
  PPAS2: Serogroup Y: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup Y: >=1:8: Day 0 before dose 3 | 89.4 [81.3 to 94.8] |
  PPAS2: Serogroup Y: >=1:4: Day 30 post dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup Y: >=1:4: Day 30 post dose 3 | 100 [96.2 to 100] |
  PPAS2: Serogroup Y: >=1:8: Day 30 post dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup Y: >=1:8: Day 30 post dose 3 | 100 [96.2 to 100] |
  PPAS2: Serogroup Y: >=1:4: Day 0 before dose 4: number analyzed (Participants) | 0 | 90
  PPAS2: Serogroup Y: >=1:4: Day 0 before dose 4 |  | 100 [96.0 to 100]
  PPAS2: Serogroup Y: >=1:8: Day 0 before dose 4: number analyzed (Participants) | 0 | 90
  PPAS2: Serogroup Y: >=1:8: Day 0 before dose 4 |  | 100 [96.0 to 100]
  PPAS2: Serogroup Y: >=1:4: Day 30 post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup Y: >=1:4: Day 30 post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup Y: >=1:8: Day 30 post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup Y: >=1:8: Day 30 post dose 4 |  | 100 [95.9 to 100]

6. Secondary Outcome: Groups 1 and 2: Percentage of Participants With Vaccine Seroresponse
Description: Functional meningococcal antibody activity against serogroups A, C, W, and Y were measured in a serum bactericidal assay utilizing the hSBA. hSBA vaccine seroresponse was defined for a participant with a pre vaccination titer <1:8, the post-vaccination titer must be >=1:16 and for a participant with a pre vaccination titer >=1:8, the post-vaccination titer must be at least 4-fold greater than the pre vaccination titer. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 Post Doses 2 and 3 (4 MoA and 12 to 18 MoA)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix
Number analyzed (Participants) | 551 | 575
Percentage of participants
  PPAS1: Serogroup A: Day 30 post dose 2: number analyzed (Participants) | 507 | 504
  PPAS1: Serogroup A: Day 30 post dose 2 | 46.7 [42.3 to 51.2] | 60.9 [56.5 to 65.2]
  PPAS1: Serogroup C: Day 30 post dose 2: number analyzed (Participants) | 508 | 514
  PPAS1: Serogroup C: Day 30 post dose 2 | 97.4 [95.7 to 98.6] | 86.8 [83.5 to 89.6]
  PPAS1: Serogroup W: Day 30 post dose 2: number analyzed (Participants) | 516 | 519
  PPAS1: Serogroup W: Day 30 post dose 2 | 92.6 [90.0 to 94.7] | 88.4 [85.4 to 91.1]
  PPAS1: Serogroup Y: Day 30 post dose 2: number analyzed (Participants) | 513 | 517
  PPAS1: Serogroup Y: Day 30 post dose 2 | 87.1 [83.9 to 89.9] | 81.4 [77.8 to 84.7]
  PPAS2: Serogroup A: Day 30 post dose 3: number analyzed (Participants) | 542 | 564
  PPAS2: Serogroup A: Day 30 post dose 3 | 90.6 [87.8 to 92.9] | 91.7 [89.1 to 93.8]
  PPAS2: Serogroup C: Day 30 post dose 3: number analyzed (Participants) | 545 | 573
  PPAS2: Serogroup C: Day 30 post dose 3 | 98.7 [97.4 to 99.5] | 91.3 [88.7 to 93.5]
  PPAS2: Serogroup W: Day 30 post dose 3: number analyzed (Participants) | 545 | 572
  PPAS2: Serogroup W: Day 30 post dose 3 | 99.4 [98.4 to 99.9] | 98.4 [97.0 to 99.3]
  PPAS2: Serogroup Y: Day 30 post dose 3 | 98.7 [97.4 to 99.5] | 96.9 [95.1 to 98.1]

7. Secondary Outcome: Groups 3 and 4: Percentage of Participants With Vaccine Seroresponse
Description: as for outcome 6
Time Frame: Group 3: Day 30 Post Dose 2 (4 MoA), Day 30 Post Dose 3 (12 to 18 MoA); Group 4: D30 Post Dose 3 (6 MoA), Day 30 Post Dose 4 (12 to 18 MoA)
Population: PPAS1 was a subset of FAS1. FAS1 included subset of randomized participants who received at least 1 dose of study vaccine in primary series and had a valid post-primary series vaccination blood sample result. PPAS2 was a subset of FAS2. FAS2 included subset of randomized participants who received at least 1 dose of study vaccine at booster vaccination and had a valid post-booster vaccination blood sample result. Only participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 94 | 90
Percentage of participants
  PPAS1: Serogroup A: Day 30 post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup A: Day 30 post dose 2 | 51.7 [40.8 to 62.4] |
  PPAS1: Serogroup A: Day 30 post dose 3: number analyzed (Participants) | 0 | 87
  PPAS1: Serogroup A: Day 30 post dose 3 |  | 65.5 [54.6 to 75.4]
  PPAS1: Serogroup C: Day 30 post dose 2: number analyzed (Participants) | 93 | 0
  PPAS1: Serogroup C: Day 30 post dose 2 | 92.5 [85.1 to 96.9] |
  PPAS1: Serogroup C: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup C: Day 30 post dose 3 |  | 96.7 [90.6 to 99.3]
  PPAS1: Serogroup W: Day 30 post dose 2: number analyzed (Participants) | 94 | 0
  PPAS1: Serogroup W: Day 30 post dose 2 | 94.7 [88.0 to 98.3] |
  PPAS1: Serogroup W: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup W: Day 30 post dose 3 |  | 95.6 [89.0 to 98.8]
  PPAS1: Serogroup Y: Day 30 post dose 2: number analyzed (Participants) | 94 | 0
  PPAS1: Serogroup Y: Day 30 post dose 2 | 89.4 [81.3 to 94.8] |
  PPAS1: Serogroup Y: Day 30 post dose 3: number analyzed (Participants) | 0 | 90
  PPAS1: Serogroup Y: Day 30 post dose 3 |  | 94.4 [87.5 to 98.2]
  PPAS2: Serogroup A: Day 30 post dose 3: number analyzed (Participants) | 90 | 0
  PPAS2: Serogroup A: Day 30 post dose 3 | 77.8 [67.8 to 85.9] |
  PPAS2: Serogroup A: Day 30 post dose 4: number analyzed (Participants) | 0 | 88
  PPAS2: Serogroup A: Day 30 post dose 4 |  | 63.6 [52.7 to 73.6]
  PPAS2: Serogroup C: Day 30 post dose 3: number analyzed (Participants) | 93 | 0
  PPAS2: Serogroup C: Day 30 post dose 3 | 97.8 [92.4 to 99.7] |
  PPAS2: Serogroup C: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup C: Day 30 post dose 4 |  | 95.3 [88.5 to 98.7]
  PPAS2: Serogroup W: Day 30 post dose 3: number analyzed (Participants) | 86 | 0
  PPAS2: Serogroup W: Day 30 post dose 3 | 97.7 [91.9 to 99.7] |
  PPAS2: Serogroup W: Day 30 post dose 4: number analyzed (Participants) | 0 | 86
  PPAS2: Serogroup W: Day 30 post dose 4 |  | 89.5 [81.1 to 95.1]
  PPAS2: Serogroup Y: Day 30 post dose 3: number analyzed (Participants) | 94 | 0
  PPAS2: Serogroup Y: Day 30 post dose 3 | 91.5 [83.9 to 96.3] |
  PPAS2: Serogroup Y: Day 30 post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup Y: Day 30 post dose 4 |  | 80.9 [71.2 to 88.5]

8. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Pertussis Antibodies
Description: GMCs of anti-pertussis antibodies (pertussis toxin [PT], filamentous hemagglutinin [FHA]) were measured by electrochemiluminescent (ECL) assay.
Time Frame: Groups 1, 2 and 3: Day 0 before Dose 1 (2 MoA); Group 4: Day 0 before Dose 4 (12 to 18 MoA)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 520 | 521 | 95 | 90
Titer
  PPAS1: Anti-PT: Day 0 before dose 1: number analyzed (Participants) | 520 | 521 | 95 | 0
  PPAS1: Anti-PT: Day 0 before dose 1 | 2.97 [2.68 to 3.29] | 2.61 [2.38 to 2.87] | 11.0 [8.74 to 14.0] |
  PPAS1: Anti-FHA: Day 0 before dose 1: number analyzed (Participants) | 520 | 521 | 95 | 0
  PPAS1: Anti-FHA: Day 0 before dose 1 | 10.8 [9.73 to 12.1] | 10.1 [9.10 to 11.2] | 55.6 [42.4 to 73.0] |
  PPAS2: Anti-PT: Day 0 before dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  PPAS2: Anti-PT: Day 0 before dose 4 |  |  |  | 10.7 [8.82 to 13.1]
  PPAS2: Anti-FHA: Day 0 before dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  PPAS2: Anti-FHA: Day 0 before dose 4 |  |  |  | 30.3 [25.0 to 36.7]

9. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Hexavalent Vaccines
Description: GMCs of hexavalent vaccines were measured as: anti-diphtheria, anti-tetanus, anti-pertussis antibodies (PT, FHA) by ECL assay, anti-hepatitis antibodies (anti-Hepatitis B surface antigen [HBsAg]) by the commercially available VITROS ECi/ECiQ, anti-poliovirus types 1, 2, and 3 by neutralization assay and anti-Haemophilus influenzae type b (anti-polyribosylribitol phosphate [PRP]) by Farr-type radioimmunoassay (RIA).
Time Frame: Groups 1, 2 and 3: Day 30 Post Doses 2 and 3 (4 MoA and 12 to 18 MoA); Day 0 Before Dose 3 (12 to 18 MoA); Group 4: Day 30 Post Dose 4 (12 to 18 MoA)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 555 | 583 | 96 | 90
Titer
  PPAS1: Anti-diphtheria: Day 30 after dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-diphtheria: Day 30 after dose 2 | 0.523 [0.474 to 0.578] | 0.489 [0.443 to 0.541] | 0.563 [0.458 to 0.691] |
  PPAS1: Anti-tetanus: Day 30 after dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-tetanus: Day 30 after dose 2 | 1.10 [1.02 to 1.18] | 1.13 [1.05 to 1.22] | 0.931 [0.788 to 1.10] |
  PPAS1: Anti-PT: Day 30 after dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-PT: Day 30 after dose 2 | 64.9 [61.4 to 68.7] | 68.1 [64.5 to 72.0] | 50.0 [43.2 to 58.0] |
  PPAS1: Anti-FHA: Day 30 after dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-FHA: Day 30 after dose 2 | 92.4 [87.3 to 97.8] | 96.6 [90.8 to 103] | 125 [109 to 144] |
  PPAS1: Anti-HBsAg: Day 30 after dose 2: number analyzed (Participants) | 505 | 510 | 92 | 0
  PPAS1: Anti-HBsAg: Day 30 after dose 2 | 369 [323 to 421] | 345 [303 to 393] | 218 [147 to 322] |
  PPAS1: Anti-polio 1: Day 30 after dose 2: number analyzed (Participants) | 486 | 489 | 83 | 0
  PPAS1: Anti-polio 1: Day 30 after dose 2 | 47.1 [40.1 to 55.3] | 43.5 [37.0 to 51.2] | 362 [260 to 504] |
  PPAS1: Anti-polio 2: Day 30 after dose 2: number analyzed (Participants) | 482 | 485 | 79 | 0
  PPAS1: Anti-polio 2: Day 30 after dose 2 | 139 [117 to 167] | 143 [120 to 171] | 618 [429 to 890] |
  PPAS1: Anti-polio 3: Day 30 after dose 2: number analyzed (Participants) | 488 | 492 | 82 | 0
  PPAS1: Anti-polio 3: Day 30 after dose 2 | 133 [112 to 157] | 145 [123 to 172] | 584 [419 to 814] |
  PPAS1: Anti-PRP: Day 30 after dose 2: number analyzed (Participants) | 517 | 521 | 96 | 0
  PPAS1: Anti-PRP: Day 30 after dose 2 | 0.376 [0.326 to 0.435] | 0.435 [0.379 to 0.499] | 0.725 [0.492 to 1.07] |
  PPAS2: Anti-diphtheria: Day 0 before dose 3: number analyzed (Participants) | 542 | 569 | 91 | 0
  PPAS2: Anti-diphtheria: Day 0 before dose 3 | 0.086 [0.079 to 0.095] | 0.080 [0.073 to 0.087] | 0.094 [0.076 to 0.116] |
  PPAS2: Anti-diphtheria: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-diphtheria: Day 30 after dose 3 | 1.82 [1.69 to 1.96] | 1.69 [1.57 to 1.81] | 2.71 [2.36 to 3.11] |
  PPAS2: Anti-diphtheria: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-diphtheria: Day 30 after dose 4 |  |  |  | 3.26 [2.88 to 3.69]
  PPAS2: Anti-tetanus: Day 0 before dose 3: number analyzed (Participants) | 542 | 571 | 92 | 0
  PPAS2: Anti-tetanus: Day 0 before dose 3 | 0.362 [0.336 to 0.391] | 0.424 [0.397 to 0.453] | 0.218 [0.180 to 0.264] |
  PPAS2: Anti-tetanus: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-tetanus: Day 30 after dose 3 | 6.71 [6.33 to 7.12] | 8.59 [8.13 to 9.08] | 6.02 [5.06 to 7.16] |
  PPAS2: Anti-tetanus: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-tetanus: Day 30 after dose 4 |  |  |  | 7.00 [5.99 to 8.18]
  PPAS2: Anti-PT: Day 0 before dose 3: number analyzed (Participants) | 542 | 571 | 92 | 0
  PPAS2: Anti-PT: Day 0 before dose 3 | 14.8 [13.8 to 15.8] | 14.6 [13.7 to 15.6] | 10.4 [8.99 to 12.0] |
  PPAS2: Anti-PT: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-PT: Day 30 after dose 3 | 111 [105 to 118] | 109 [104 to 115] | 79.2 [66.2 to 94.6] |
  PPAS2: Anti-PT: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-PT: Day 30 after dose 4 |  |  |  | 80.9 [68.2 to 95.9]
  PPAS2: Anti-FHA: Day 0 before dose 3: number analyzed (Participants) | 542 | 571 | 92 | 0
  PPAS2: Anti-FHA: Day 0 before dose 3 | 38.4 [35.8 to 41.2] | 38.1 [35.5 to 40.8] | 30.6 [26.0 to 36.0] |
  PPAS2: Anti-FHA: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-FHA: Day 30 after dose 3 | 177 [167 to 187] | 184 [173 to 195] | 168 [142 to 200] |
  PPAS2: Anti-FHA: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-FHA: Day 30 after dose 4 |  |  |  | 181 [151 to 217]
  PPAS2: Anti-HBsAg: Day 0 before dose 3: number analyzed (Participants) | 535 | 565 | 91 | 0
  PPAS2: Anti-HBsAg: Day 0 before dose 3 | 53.0 [45.5 to 61.8] | 48.8 [42.1 to 56.5] | 26.0 [17.6 to 38.2] |
  PPAS2: Anti-HBsAg: Day 30 after dose 3: number analyzed (Participants) | 546 | 571 | 90 | 0
  PPAS2: Anti-HBsAg: Day 30 after dose 3 | 2273 [1927 to 2681] | 2158 [1852 to 2515] | 1117 [666 to 1872] |
  PPAS2: Anti-HBsAg: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 86
  PPAS2: Anti-HBsAg: Day 30 after dose 4 |  |  |  | 1144 [648 to 2020]
  PPAS2: Anti-polio 1: Day 0 before dose 3: number analyzed (Participants) | 526 | 559 | 89 | 0
  PPAS2: Anti-polio 1: Day 0 before dose 3 | 14.5 [12.7 to 16.5] | 13.6 [12.0 to 15.4] | 55.2 [40.8 to 74.6] |
  PPAS2: Anti-polio 1: Day 30 after dose 3: number analyzed (Participants) | 533 | 553 | 86 | 0
  PPAS2: Anti-polio 1: Day 30 after dose 3 | 1099 [980 to 1233] | 994 [883 to 1119] | 1538 [1212 to 1952] |
  PPAS2: Anti-polio 1: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 87
  PPAS2: Anti-polio 1: Day 30 after dose 4 |  |  |  | 1625 [1291 to 2047]
  PPAS2: Anti-polio 2: Day 0 before dose 3: number analyzed (Participants) | 528 | 560 | 88 | 0
  PPAS2: Anti-polio 2: Day 0 before dose 3 | 33.2 [28.7 to 38.4] | 33.1 [28.8 to 37.9] | 85.3 [63.9 to 114] |
  PPAS2: Anti-polio 2: Day 30 after dose 3: number analyzed (Participants) | 530 | 554 | 87 | 0
  PPAS2: Anti-polio 2: Day 30 after dose 3 | 2214 [1982 to 2472] | 2146 [1937 to 2379] | 3549 [2846 to 4425] |
  PPAS2: Anti-polio 2: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 87
  PPAS2: Anti-polio 2: Day 30 after dose 4 |  |  |  | 3858 [3001 to 4960]
  PPAS2: Anti-polio 3: Day 0 before dose 3: number analyzed (Participants) | 529 | 560 | 89 | 0
  PPAS2: Anti-polio 3: Day 0 before dose 3 | 19.7 [17.1 to 22.6] | 18.4 [16.0 to 21.1] | 37.7 [27.6 to 51.5] |
  PPAS2: Anti-polio 3: Day 30 after dose 3: number analyzed (Participants) | 531 | 557 | 87 | 0
  PPAS2: Anti-polio 3: Day 30 after dose 3 | 1595 [1393 to 1827] | 1533 [1361 to 1728] | 2431 [1897 to 3115] |
  PPAS2: Anti-polio 3: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 87
  PPAS2: Anti-polio 3: Day 30 after dose 4 |  |  |  | 3397 [2567 to 4495]
  PPAS2: Anti-PRP: Day 0 before dose 3: number analyzed (Participants) | 545 | 571 | 93 | 0
  PPAS2: Anti-PRP: Day 0 before dose 3 | 0.201 [0.176 to 0.230] | 0.224 [0.197 to 0.255] | 0.244 [0.174 to 0.343] |
  PPAS2: Anti-PRP: Day 30 after dose 3: number analyzed (Participants) | 555 | 583 | 91 | 0
  PPAS2: Anti-PRP: Day 30 after dose 3 | 9.42 [8.31 to 10.7] | 11.5 [10.3 to 12.9] | 16.1 [11.9 to 21.6] |
  PPAS2: Anti-PRP: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  PPAS2: Anti-PRP: Day 30 after dose 4 |  |  |  | 16.1 [12.1 to 21.6]

10. Secondary Outcome: Percentage of Participants With Response Rate for Anti-Diphtheria, Anti-Tetanus, Anti-Poliovirus Types 1, 2, and 3, Anti-Haemophilus Influenzae Type b (Anti-PRP)
Description: GMCs of anti-diphtheria, anti-tetanus, anti-poliovirus types 1, 2, and 3, anti-haemophilus influenzae type b (anti-PRP) vaccines were measured as: anti-diphtheria, anti-tetanus by ECL assay, anti-poliovirus types 1, 2, and 3 by neutralization assay and anti-Haemophilus influenzae type b (anti-PRP) by Farr-type RIA. Response rate was defined as percentage of participants who achieved: anti diphtheria and anti-tetanus antibody concentrations >=0.01 international units (IU)/milliliter (mL), >=0.1 IU/mL and >=1.0 IU/mL; anti-poliovirus types 1, 2, and 3 antibody titers >=1:8; anti-PRP antibody concentrations >=0.15 microgram (mcg)/mL and >=1 mcg/mL. Percentages are rounded off to the tenth decimal place.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 555 | 583 | 96 | 90
Percentage of participants
  PPAS1: Anti-diphtheria: >=0.01 IU/mL: Day 30 post dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-diphtheria: >=0.01 IU/mL: Day 30 post dose 2 | 100 [99.3 to 100] | 99.8 [98.9 to 100] | 100 [96.1 to 100] |
  PPAS1: Anti-diphtheria: >=0.1 IU/mL: Day 30 post dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-diphtheria: >=0.1 IU/mL: Day 30 post dose 2 | 90.5 [87.6 to 92.9] | 89.6 [86.7 to 92.1] | 94.6 [87.9 to 98.2] |
  PPAS1: Anti-diphtheria: >=1.0 IU/mL: Day 30 post dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-diphtheria: >=1.0 IU/mL: Day 30 post dose 2 | 32.7 [28.6 to 36.9] | 32.5 [28.5 to 36.7] | 33.3 [23.9 to 43.9] |
  PPAS1: Anti-tetanus: >=0.01 IU/mL: Day 30 post dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-tetanus: >=0.01 IU/mL: Day 30 post dose 2 | 100 [99.3 to 100] | 100 [99.3 to 100] | 100 [96.1 to 100] |
  PPAS1: Anti-tetanus: >=0.1 IU/mL: Day 30 post dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-tetanus: >=0.1 IU/mL: Day 30 post dose 2 | 100 [99.3 to 100] | 99.8 [98.9 to 100] | 100 [96.1 to 100] |
  PPAS1: Anti-tetanus: >=1.0 IU/mL: Day 30 post dose 2: number analyzed (Participants) | 514 | 520 | 93 | 0
  PPAS1: Anti-tetanus: >=1.0 IU/mL: Day 30 post dose 2 | 53.3 [48.9 to 57.7] | 56.3 [52.0 to 60.7] | 44.1 [33.8 to 54.8] |
  PPAS1: Anti-polio 1: >=1:8: Day 30 post dose 2: number analyzed (Participants) | 486 | 489 | 83 | 0
  PPAS1: Anti-polio 1: >=1:8: Day 30 post dose 2 | 87.0 [83.7 to 89.9] | 83.2 [79.6 to 86.4] | 98.8 [93.5 to 100] |
  PPAS1: Anti-polio 2:>=1:8: Day 30 post dose 2: number analyzed (Participants) | 482 | 485 | 79 | 0
  PPAS1: Anti-polio 2:>=1:8: Day 30 post dose 2 | 97.5 [95.7 to 98.7] | 98.6 [97.0 to 99.4] | 100 [95.4 to 100] |
  PPAS1: Anti-polio 3:>=1:8: Day 30 post dose 2: number analyzed (Participants) | 488 | 492 | 82 | 0
  PPAS1: Anti-polio 3:>=1:8: Day 30 post dose 2 | 95.9 [93.7 to 97.5] | 96.1 [94.0 to 97.7] | 98.8 [93.4 to 100] |
  PPAS1: Anti-PRP: >=0.15 mcg/mL: Day 30 post dose 2: number analyzed (Participants) | 517 | 521 | 96 | 0
  PPAS1: Anti-PRP: >=0.15 mcg/mL: Day 30 post dose 2 | 71.8 [67.7 to 75.6] | 74.9 [70.9 to 78.5] | 78.1 [68.5 to 85.9] |
  PPAS1: Anti-PRP: >=1 mcg/mL: Day 30 post dose 2: number analyzed (Participants) | 517 | 521 | 96 | 0
  PPAS1: Anti-PRP: >=1 mcg/mL: Day 30 post dose 2 | 24.2 [20.5 to 28.1] | 27.3 [23.5 to 31.3] | 39.6 [29.7 to 50.1] |
  PPAS2: Anti-diphtheria: >=0.01 IU/mL: Day 0 before dose 3: number analyzed (Participants) | 542 | 569 | 91 | 0
  PPAS2: Anti-diphtheria: >=0.01 IU/mL: Day 0 before dose 3 | 98.2 [96.6 to 99.1] | 98.6 [97.2 to 99.4] | 97.8 [92.3 to 99.7] |
  PPAS2: Anti-diphtheria: >=0.01 IU/mL: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-diphtheria: >=0.01 IU/mL: Day 30 after dose 3 | 100 [99.3 to 100] | 100 [99.4 to 100] | 100 [96.1 to 100] |
  PPAS2: Anti-diphtheria: >=0.01 IU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-diphtheria: >=0.01 IU/mL: Day 30 after dose 4 |  |  |  | 100 [95.9 to 100]
  PPAS2: Anti-diphtheria: >=0.1 IU/mL: Day 0 before dose 3: number analyzed (Participants) | 542 | 569 | 91 | 0
  PPAS2: Anti-diphtheria: >=0.1 IU/mL: Day 0 before dose 3 | 48.2 [43.9 to 52.5] | 41.3 [37.2 to 45.5] | 47.3 [36.7 to 58.0] |
  PPAS2: Anti-diphtheria: >=0.1 IU/mL: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-diphtheria: >=0.1 IU/mL: Day 30 after dose 3 | 99.6 [98.7 to 100] | 99.8 [99.0 to 100] | 100 [96.1 to 100] |
  PPAS2: Anti-diphtheria: >=0.1 IU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-diphtheria: >=0.1 IU/mL: Day 30 after dose 4 |  |  |  | 100 [95.9 to 100]
  PPAS2: Anti-diphtheria: >=1.0 IU/mL: Day 0 before dose 3: number analyzed (Participants) | 542 | 569 | 91 | 0
  PPAS2: Anti-diphtheria: >=1.0 IU/mL: Day 0 before dose 3 | 1.1 [0.4 to 2.4] | 0.7 [0.2 to 1.8] | 0 [0 to 4.0] |
  PPAS2: Anti-diphtheria: >=1.0 IU/mL: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-diphtheria: >=1.0 IU/mL: Day 30 after dose 3 | 75.5 [71.7 to 79.0] | 72.4 [68.6 to 76.1] | 92.4 [84.9 to 96.9] |
  PPAS2: Anti-diphtheria: >=1.0 IU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-diphtheria: >=1.0 IU/mL: Day 30 after dose 4 |  |  |  | 100 [95.9 to 100]
  PPAS2: Anti-tetanus: >=0.01 IU/mL: Day 0 before dose 3: number analyzed (Participants) | 542 | 571 | 92 | 0
  PPAS2: Anti-tetanus: >=0.01 IU/mL: Day 0 before dose 3 | 100 [99.3 to 100] | 100 [99.4 to 100] | 100 [96.1 to 100] |
  PPAS2: Anti-tetanus: >=0.01 IU/mL: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-tetanus: >=0.01 IU/mL: Day 30 after dose 3 | 100 [99.3 to 100] | 100 [99.4 to 100] | 100 [96.1 to 100] |
  PPAS2: Anti-tetanus: >=0.01 IU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-tetanus: >=0.01 IU/mL: Day 30 after dose 4 |  |  |  | 100 [95.9 to 100]
  PPAS2: Anti- tetanus: >=0.1 IU/mL: Day 0 before dose 3: number analyzed (Participants) | 542 | 571 | 92 | 0
  PPAS2: Anti- tetanus: >=0.1 IU/mL: Day 0 before dose 3 | 94.1 [91.8 to 95.9] | 97.4 [95.7 to 98.5] | 83.7 [74.5 to 90.6] |
  PPAS2: Anti-tetanus: >=0.1 IU/mL: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-tetanus: >=0.1 IU/mL: Day 30 after dose 3 | 100 [99.3 to 100] | 100 [99.4 to 100] | 100 [96.1 to 100] |
  PPAS2: Anti-tetanus: >=0.1 IU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-tetanus: >=0.1 IU/mL: Day 30 after dose 4 |  |  |  | 100 [95.9 to 100]
  PPAS2: Anti-tetanus: >=1.0 IU/mL: Day 0 before dose 3: number analyzed (Participants) | 542 | 571 | 92 | 0
  PPAS2: Anti-tetanus: >=1.0 IU/mL: Day 0 before dose 3 | 10.7 [8.2 to 13.6] | 14.7 [11.9 to 17.9] | 6.5 [2.4 to 13.7] |
  PPAS2: Anti-tetanus: >=1.0 IU/mL: Day 30 after dose 3: number analyzed (Participants) | 551 | 577 | 92 | 0
  PPAS2: Anti-tetanus: >=1.0 IU/mL: Day 30 after dose 3 | 99.6 [98.7 to 100] | 99.7 [98.8 to 100] | 96.7 [90.8 to 99.3] |
  PPAS2: Anti-tetanus: >=1.0 IU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-tetanus: >=1.0 IU/mL: Day 30 after dose 4 |  |  |  | 98.9 [93.9 to 100]
  PPAS2: Anti-polio 1: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 526 | 559 | 89 | 0
  PPAS2: Anti-polio 1: >=1:8: Day 0 before dose 3 | 64.4 [60.2 to 68.5] | 63.7 [59.5 to 67.7] | 93.3 [85.9 to 97.5] |
  PPAS2: Anti-polio 1: >=1:8: Day 30 after dose 3: number analyzed (Participants) | 533 | 553 | 86 | 0
  PPAS2: Anti-polio 1: >=1:8: Day 30 after dose 3 | 99.8 [99.0 to 100] | 98.9 [97.7 to 99.6] | 100 [95.8 to 100] |
  PPAS2: Anti-polio 1: >=1:8: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 87
  PPAS2: Anti-polio 1: >=1:8: Day 30 after dose 4 |  |  |  | 100 [95.8 to 100]
  PPAS2: Anti-polio 2: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 528 | 560 | 88 | 0
  PPAS2: Anti-polio 2: >=1:8: Day 0 before dose 3 | 79.5 [75.8 to 82.9] | 80.9 [77.4 to 84.1] | 95.5 [88.8 to 98.7] |
  PPAS2: Anti-polio 2: >=1:8: Day 30 after dose 3: number analyzed (Participants) | 530 | 554 | 87 | 0
  PPAS2: Anti-polio 2: >=1:8: Day 30 after dose 3 | 100 [99.3 to 100] | 100 [99.3 to 100] | 100 [95.8 to 100] |
  PPAS2: Anti-polio 2: >=1:8: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 87
  PPAS2: Anti-polio 2: >=1:8: Day 30 after dose 4 |  |  |  | 100 [95.8 to 100]
  PPAS2: Anti-polio 3: >=1:8: Day 0 before dose 3: number analyzed (Participants) | 529 | 560 | 89 | 0
  PPAS2: Anti-polio 3: >=1:8: Day 0 before dose 3 | 68.6 [64.5 to 72.6] | 65.7 [61.6 to 69.6] | 84.3 [75.0 to 91.1] |
  PPAS2: Anti-polio 3: >=1:8: Day 30 after dose 3: number analyzed (Participants) | 531 | 557 | 87 | 0
  PPAS2: Anti-polio 3: >=1:8: Day 30 after dose 3 | 99.2 [98.1 to 99.8] | 99.8 [99.0 to 100] | 100 [95.8 to 100] |
  PPAS2: Anti-polio 3: >=1:8: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 87
  PPAS2: Anti-polio 3: >=1:8: Day 30 after dose 4 |  |  |  | 100 [95.8 to 100]
  PPAS2: Anti-PRP: >=0.15 mcg/mL: Day 0 before dose 3: number analyzed (Participants) | 545 | 571 | 93 | 0
  PPAS2: Anti-PRP: >=0.15 mcg/mL: Day 0 before dose 3 | 56.5 [52.2 to 60.7] | 60.4 [56.3 to 64.5] | 60.2 [49.5 to 70.2] |
  PPAS2: Anti-PRP: >=0.15 mcg/mL: Day 30 after dose 3: number analyzed (Participants) | 555 | 583 | 91 | 0
  PPAS2: Anti-PRP: >=0.15 mcg/mL: Day 30 after dose 3 | 98.2 [96.7 to 99.1] | 98.8 [97.5 to 99.5] | 100 [96.0 to 100] |
  PPAS2: Anti-PRP: >=0.15 mcg/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  PPAS2: Anti-PRP: >=0.15 mcg/mL: Day 30 after dose 4 |  |  |  | 100 [96.0 to 100]
  PPAS2: Anti-PRP: >=1 mcg/mL: Day 0 before dose 3: number analyzed (Participants) | 545 | 571 | 93 | 0
  PPAS2: Anti-PRP: >=1 mcg/mL: Day 0 before dose 3 | 13.9 [11.1 to 17.1] | 14.9 [12.1 to 18.1] | 15.1 [8.5 to 24.0] |
  PPAS2: Anti-PRP: >=1 mcg/mL: Day 30 after dose 3: number analyzed (Participants) | 555 | 583 | 91 | 0
  PPAS2: Anti-PRP: >=1 mcg/mL: Day 30 after dose 3 | 91.5 [88.9 to 93.7] | 94.9 [92.7 to 96.5] | 97.8 [92.3 to 99.7] |
  PPAS2: Anti-PRP: >=1 mcg/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  PPAS2: Anti-PRP: >=1 mcg/mL: Day 30 after dose 4 |  |  |  | 96.7 [90.6 to 99.3]

11. Secondary Outcome: Percentage of Participants Who Achieved Vaccine Seroresponse for Anti-Pertussis Antibodies
Description: GMCs of anti-pertussis antibodies (PT, FHA) were measured by ECL assay. The pertussis vaccine seroresponse for anti-PT and anti-FHA was defined as: For groups 1, 2, and 3, 30 days after dose 2 in infancy as if the pre-primary vaccination concentration is <4 × lower limit of quantification (LLOQ), post-primary vaccination concentration >=4 × LLOQ, if the pre-primary vaccination concentration is >=4 ×LLOQ, post-primary vaccination concentration >=pre-primary vaccination concentration; and for Groups 1, 2, and 3, before and 30 days after the dose 3 and for group 4, before and 30 days after the dose 4 as if the pre-booster vaccination concentration is <4 × LLOQ, post-booster vaccination concentration >=4 × pre-booster concentration, if the pre-booster vaccination concentration is >=4 × LLOQ, post-booster vaccination concentration >=2 × pre-booster concentration. Percentages are rounded off to the tenth decimal place.
Time Frame: Groups 1, 2 and 3: Day 30 Post Doses 2 and 3 (4 MoA and 12 to 18 MoA); Group 4: Day 30 Post Dose 4 (12 to 18 MoA)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 533 | 565 | 92 | 89
Percentage of participants
  PPAS1: Anti-PT: Day 30 post dose 2: number analyzed (Participants) | 512 | 518 | 92 | 0
  PPAS1: Anti-PT: Day 30 post dose 2 | 94.5 [92.2 to 96.3] | 97.9 [96.2 to 98.9] | 82.6 [73.3 to 89.7] |
  PPAS1: Anti-FHA: Day 30 post dose 2: number analyzed (Participants) | 512 | 518 | 92 | 0
  PPAS1: Anti-FHA: Day 30 post dose 2 | 89.6 [86.7 to 92.1] | 91.5 [88.8 to 93.8] | 62.0 [51.2 to 71.9] |
  PPAS2: Anti-PT: Day 30 post dose 3: number analyzed (Participants) | 533 | 565 | 90 | 0
  PPAS2: Anti-PT: Day 30 post dose 3 | 97.0 [95.2 to 98.3] | 97.0 [95.2 to 98.2] | 93.3 [86.1 to 97.5] |
  PPAS2: Anti-PT: Day 30 post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-PT: Day 30 post dose 4 |  |  |  | 88.8 [80.3 to 94.5]
  PPAS2: Anti-FHA: Day 30 post dose 3: number analyzed (Participants) | 533 | 565 | 90 | 0
  PPAS2: Anti-FHA: Day 30 post dose 3 | 89.1 [86.2 to 91.6] | 90.1 [87.3 to 92.4] | 92.2 [84.6 to 96.8] |
  PPAS2: Anti-FHA: Day 30 post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 89
  PPAS2: Anti-FHA: Day 30 post dose 4 |  |  |  | 91.0 [83.1 to 96.0]

12. Secondary Outcome: Percentage of Participants Who Achieved Anti-Hepatitis B Antibody Concentrations >=10 and >=100 Milli-International Units (mIU)/mL
Description: GMCs of anti-hepatitis antibodies (anti-HBsAg) was measured by the commercially available VITROS ECi/ECiQ. Response rate for anti-HBsAg was defined as percentage of participants who achieved anti-HBsAg antibody concentrations >=10 mIU/mL and >=100 mIU/mL. Percentages are rounded off to the tenth decimal place.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 546 | 571 | 92 | 90
Percentage of participants
  PPAS1: Anti-HBsAg: >=10 mIU/mL: Day 30 post dose 2: number analyzed (Participants) | 505 | 510 | 92 | 0
  PPAS1: Anti-HBsAg: >=10 mIU/mL: Day 30 post dose 2 | 96.4 [94.4 to 97.9] | 97.8 [96.2 to 98.9] | 92.4 [84.9 to 96.9] |
  PPAS1: Anti-HBsAg: >=100 mIU/mL: Day 30 post dose 2: number analyzed (Participants) | 505 | 510 | 92 | 0
  PPAS1: Anti-HBsAg: >=100 mIU/mL: Day 30 post dose 2 | 85.7 [82.4 to 88.7] | 81.8 [78.1 to 85.0] | 72.8 [62.6 to 81.6] |
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 0 before dose 3: number analyzed (Participants) | 535 | 565 | 91 | 0
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 0 before dose 3 | 81.5 [77.9 to 84.7] | 79.5 [75.9 to 82.7] | 65.9 [55.3 to 75.5] |
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 30 after dose 3: number analyzed (Participants) | 546 | 571 | 90 | 0
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 30 after dose 3 | 98.0 [96.4 to 99.0] | 98.6 [97.3 to 99.4] | 94.4 [87.5 to 98.2] |
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 0 before dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 0 before dose 4 |  |  |  | 64.4 [53.7 to 74.3]
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 86
  PPAS2: Anti-HBsAg: >=10 mIU/mL: Day 30 after dose 4 |  |  |  | 91.9 [83.9 to 96.7]
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 0 before dose 3: number analyzed (Participants) | 535 | 565 | 91 | 0
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 0 before dose 3 | 38.7 [34.5 to 43.0] | 35.4 [31.5 to 39.5] | 26.4 [17.7 to 36.7] |
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 30 after dose 3: number analyzed (Participants) | 546 | 571 | 90 | 0
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 30 after dose 3 | 93.4 [91.0 to 95.3] | 93.5 [91.2 to 95.4] | 80.0 [70.2 to 87.7] |
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 0 before dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 0 before dose 4 |  |  |  | 27.8 [18.9 to 38.2]
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 30 after dose 4: number analyzed (Participants) | 0 | 0 | 0 | 86
  PPAS2: Anti-HBsAg: >=100 mIU/mL: Day 30 after dose 4 |  |  |  | 83.7 [74.2 to 90.8]

13. Secondary Outcome: Groups 1 and 2: Geometric Mean Concentrations (GMCs) of Pneumococcal Conjugate Vaccine (10-Valent, Adsorbed) (PCV10) Vaccine
Description: GMCs of anti-pneumococcal antibodies was assessed by pneumococcal capsular polysaccharide (PnPS) Immunoglobulin G (IgG) ECL assay which was used to quantitate the amount of anti-streptococcus pneumoniae PS (serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F) antibodies in human serum.
Time Frame: At 30 days post Dose 2 (4 MoA) and Dose 3 (12 to 18 MoA)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix
Number analyzed (Participants) | 545 | 569
Titer
  PPAS1: Serogroup 1: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 1 | 1.68 [1.52 to 1.84] | 1.71 [1.56 to 1.87]
  PPAS1: Serogroup 4: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 4 | 1.97 [1.83 to 2.12] | 2.06 [1.91 to 2.23]
  PPAS1: Serogroup 5: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 5 | 1.08 [0.991 to 1.17] | 1.10 [1.01 to 1.19]
  PPAS1: Serogroup 6B: number analyzed (Participants) | 505 | 511
  PPAS1: Serogroup 6B | 0.600 [0.534 to 0.675] | 0.660 [0.586 to 0.742]
  PPAS1: Serogroup 7F: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 7F | 2.03 [1.89 to 2.17] | 2.20 [2.05 to 2.37]
  PPAS1: Serogroup 9V: number analyzed (Participants) | 504 | 512
  PPAS1: Serogroup 9V | 1.67 [1.54 to 1.81] | 1.81 [1.67 to 1.96]
  PPAS1: Serogroup 14: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 14 | 5.92 [5.41 to 6.48] | 5.97 [5.44 to 6.55]
  PPAS1: Serogroup 18C: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 18C | 0.680 [0.618 to 0.748] | 0.796 [0.722 to 0.879]
  PPAS1: Serogroup 19F: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 19F | 1.59 [1.39 to 1.82] | 1.45 [1.26 to 1.66]
  PPAS1: Serogroup 23F: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 23F | 0.830 [0.746 to 0.924] | 0.869 [0.785 to 0.961]
  PPAS2: Serogroup 1 | 4.71 [4.32 to 5.13] | 4.54 [4.18 to 4.94]
  PPAS2: Serogroup 4 | 3.61 [3.37 to 3.86] | 3.19 [2.99 to 3.41]
  PPAS2: Serogroup 5: number analyzed (Participants) | 544 | 569
  PPAS2: Serogroup 5 | 2.21 [2.05 to 2.39] | 2.05 [1.90 to 2.20]
  PPAS2: Serogroup 6B | 4.21 [3.89 to 4.55] | 4.36 [4.04 to 4.71]
  PPAS2: Serogroup 7F: number analyzed (Participants) | 545 | 568
  PPAS2: Serogroup 7F | 2.91 [2.73 to 3.10] | 2.89 [2.70 to 3.10]
  PPAS2: Serogroup 9V | 4.08 [3.80 to 4.38] | 4.17 [3.89 to 4.47]
  PPAS2: Serogroup 14: number analyzed (Participants) | 544 | 568
  PPAS2: Serogroup 14 | 9.07 [8.44 to 9.75] | 7.89 [7.25 to 8.59]
  PPAS2: Serogroup 18C | 2.12 [1.99 to 2.26] | 2.17 [2.03 to 2.33]
  PPAS2: Serogroup 19F | 9.03 [8.32 to 9.81] | 8.41 [7.76 to 9.12]
  PPAS2: Serogroup 23F | 2.24 [2.10 to 2.40] | 2.04 [1.90 to 2.18]

14. Secondary Outcome: Groups 3 and 4: Geometric Mean Concentrations (GMCs) of Pneumococcal Conjugate Vaccine (13-Valent, Adsorbed) (PCV13) Vaccine
Description: GMCs of anti-pneumococcal antibodies was assessed by PnPS IgG ECL assay which was used to quantitate the amount of anti-streptococcus pneumoniae PS (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) antibodies in human serum.
Time Frame: Group 3: At 30 days post Dose 2 (4 MoA) and Dose 3 (12 to 18 MoA); Group 4: At 30 days post Dose 4 (12 to 18 MoA)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 91 | 89
Titer
  PPAS1: Serogroup 1: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 1: 30 days post dose 2 | 1.47 [1.16 to 1.87] |
  PPAS1: Serogroup 3: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 3: 30 days post dose 2 | 0.658 [0.554 to 0.781] |
  PPAS1: Serogroup 4: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 4: 30 days post dose 2 | 1.73 [1.42 to 2.12] |
  PPAS1: Serogroup 5: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 5: 30 days post dose 2 | 0.803 [0.617 to 1.04] |
  PPAS1: Serogroup 6A: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 6A: 30 days post dose 2 | 1.65 [1.24 to 2.19] |
  PPAS1: Serogroup 6B: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 6B: 30 days post dose 2 | 0.275 [0.205 to 0.368] |
  PPAS1: Serogroup 7F: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 7F: 30 days post dose 2 | 3.04 [2.59 to 3.57] |
  PPAS1: Serogroup 9V: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 9V: 30 days post dose 2 | 1.25 [0.987 to 1.59] |
  PPAS1: Serogroup 14: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 14: 30 days post dose 2 | 5.88 [4.31 to 8.01] |
  PPAS1: Serogroup 18C: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 18C: 30 days post dose 2 | 1.65 [1.30 to 2.10] |
  PPAS1: Serogroup 19A: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 19A: 30 days post dose 2 | 2.17 [1.67 to 2.80] |
  PPAS1: Serogroup 19F: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 19F: 30 days post dose 2 | 5.73 [4.64 to 7.08] |
  PPAS1: Serogroup 23F: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 23F: 30 days post dose 2 | 0.722 [0.552 to 0.945] |
  PPAS2: Serogroup 1: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 1: 30 days post dose 3 | 5.32 [4.41 to 6.42] |
  PPAS2: Serogroup 1: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 1: 30 days post dose 4 |  | 5.47 [4.66 to 6.42]
  PPAS2: Serogroup 3: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 3: 30 days post dose 3 | 1.13 [0.945 to 1.35] |
  PPAS2: Serogroup 3: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 3: 30 days post dose 4 |  | 1.21 [0.982 to 1.50]
  PPAS2: Serogroup 4: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 4: 30 days post dose 3 | 3.99 [3.43 to 4.64] |
  PPAS2: Serogroup 4: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 4: 30 days post dose 4 |  | 3.97 [3.35 to 4.70]
  PPAS2: Serogroup 5: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 5: 30 days post dose 3 | 3.33 [2.75 to 4.03] |
  PPAS2: Serogroup 5: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 5: 30 days post dose 4 |  | 3.95 [3.36 to 4.65]
  PPAS2: Serogroup 6A: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 6A: 30 days post dose 3 | 12.9 [10.9 to 15.4] |
  PPAS2: Serogroup 6A: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 6A: 30 days post dose 4 |  | 14.3 [12.2 to 16.8]
  PPAS2: Serogroup 6B: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 6B: 30 days post dose 3 | 7.01 [5.38 to 9.13] |
  PPAS2: Serogroup 6B: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 6B: 30 days post dose 4 |  | 9.41 [7.86 to 11.3]
  PPAS2: Serogroup 7F: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 7F: 30 days post dose 3 | 5.36 [4.56 to 6.29] |
  PPAS2: Serogroup 7F: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 7F: 30 days post dose 4 |  | 4.92 [4.20 to 5.76]
  PPAS2: Serogroup 9V: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 9V: 30 days post dose 3 | 5.12 [4.26 to 6.17] |
  PPAS2: Serogroup 9V: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 9V: 30 days post dose 4 |  | 5.40 [4.65 to 6.26]
  PPAS2: Serogroup 14: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 14: 30 days post dose 3 | 14.8 [12.2 to 18.1] |
  PPAS2: Serogroup 14: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 14: 30 days post dose 4 |  | 14.7 [12.1 to 17.9]
  PPAS2: Serogroup 18C: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 18C: 30 days post dose 3 | 3.18 [2.70 to 3.76] |
  PPAS2: Serogroup 18C: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 18C: 30 days post dose 4 |  | 3.48 [3.00 to 4.03]
  PPAS2: Serogroup 19A: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 19A: 30 days post dose 3 | 8.82 [7.25 to 10.7] |
  PPAS2: Serogroup 19A: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 19A: 30 days post dose 4 |  | 10.9 [9.26 to 12.9]
  PPAS2: Serogroup 19F: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 19F: 30 days post dose 3 | 12.1 [9.91 to 14.7] |
  PPAS2: Serogroup 19F: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 19F: 30 days post dose 4 |  | 12.2 [10.5 to 14.2]
  PPAS2: Serogroup 23F: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 23F: 30 days post dose 3 | 3.70 [3.01 to 4.55] |
  PPAS2: Serogroup 23F: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 23F: 30 days post dose 4 |  | 4.06 [3.45 to 4.76]

15. Secondary Outcome: Groups 1 and 2: Percentage of Participants With Response Rate >=0.35 mcg/mL for Pneumococcal Conjugate Vaccine (10-Valent, Adsorbed) PCV10 Vaccine
Description: GMCs of anti-pneumococcal antibodies was assessed by PnPS IgG ECL assay which was used to quantitate the amount of anti-streptococcus pneumoniae PS (serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F) antibodies in human serum. Percentages are rounded off to the tenth decimal place.
Time Frame: At 30 days post Dose 2 (4 MoA) and Dose 3 (12 to 18 MoA)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix
Number analyzed (Participants) | 545 | 569
Percentage of participants
  PPAS1: Serogroup 1: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 1 | 92.7 [90.0 to 94.8] | 93.6 [91.1 to 95.5]
  PPAS1: Serogroup 4: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 4 | 96.8 [94.9 to 98.2] | 96.7 [94.7 to 98.1]
  PPAS1: Serogroup 5: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 5 | 88.5 [85.4 to 91.2] | 90.6 [87.8 to 93.0]
  PPAS1: Serogroup 6B: number analyzed (Participants) | 505 | 511
  PPAS1: Serogroup 6B | 67.1 [62.8 to 71.2] | 69.9 [65.7 to 73.8]
  PPAS1: Serogroup 7F: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 7F | 98.8 [97.4 to 99.6] | 98.2 [96.7 to 99.2]
  PPAS1: Serogroup 9V: number analyzed (Participants) | 504 | 512
  PPAS1: Serogroup 9V | 94.6 [92.3 to 96.4] | 95.1 [92.9 to 96.8]
  PPAS1: Serogroup 14: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 14 | 97.8 [96.1 to 98.9] | 98.2 [96.7 to 99.2]
  PPAS1: Serogroup 18C: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 18C | 72.5 [68.4 to 76.3] | 77.3 [73.5 to 80.9]
  PPAS1: Serogroup 19F: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 19F | 82.2 [78.6 to 85.4] | 79.3 [75.5 to 82.7]
  PPAS1: Serogroup 23F: number analyzed (Participants) | 505 | 512
  PPAS1: Serogroup 23F | 77.8 [73.9 to 81.4] | 80.3 [76.6 to 83.6]
  PPAS2: Serogroup 1 | 99.8 [99.0 to 100] | 99.8 [99.0 to 100]
  PPAS2: Serogroup 4 | 99.8 [99.0 to 100] | 99.6 [98.7 to 100]
  PPAS2: Serogroup 5: number analyzed (Participants) | 544 | 569
  PPAS2: Serogroup 5 | 98.2 [96.6 to 99.1] | 97.7 [96.1 to 98.8]
  PPAS2: Serogroup 6B | 98.9 [97.6 to 99.6] | 99.5 [98.5 to 99.9]
  PPAS2: Serogroup 7F: number analyzed (Participants) | 545 | 568
  PPAS2: Serogroup 7F | 99.6 [98.7 to 100] | 99.3 [98.2 to 99.8]
  PPAS2: Serogroup 9V | 99.8 [99.0 to 100] | 99.8 [99.0 to 100]
  PPAS2: Serogroup 14: number analyzed (Participants) | 544 | 568
  PPAS2: Serogroup 14 | 100 [99.3 to 100] | 99.3 [98.2 to 99.8]
  PPAS2: Serogroup 18C | 99.1 [97.9 to 99.7] | 98.6 [97.2 to 99.4]
  PPAS2: Serogroup 19F | 99.3 [98.1 to 99.8] | 99.3 [98.2 to 99.8]
  PPAS2: Serogroup 23F | 98.5 [97.1 to 99.4] | 97.2 [95.5 to 98.4]

16. Secondary Outcome: Groups 3 and 4: Percentage of Participants With Response Rate >=0.35 mcg/mL for Pneumococcal Conjugate Vaccine (13-Valent, Adsorbed) PCV13 Vaccine
Description: GMCs of anti-pneumococcal antibodies was assessed by PnPS IgG ECL assay which was used to quantitate the amount of anti-streptococcus pneumoniae PS (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) antibodies in human serum. Percentages are rounded off to the tenth decimal place.
Time Frame: Group 3: At 30 days post Dose 2 (4 MoA) and Dose 3 (12 to 18 MoA); Group 4: At 30 days post Dose 4 (12 to 18 MoA)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 91 | 89
Percentage of participants
  PPAS1: Serogroup 1: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 1: 30 days post dose 2 | 89.9 [81.7 to 95.3] |
  PPAS1: Serogroup 3: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 3: 30 days post dose 2 | 82.0 [72.5 to 89.4] |
  PPAS1: Serogroup 4: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 4: 30 days post dose 2 | 96.6 [90.5 to 99.3] |
  PPAS1: Serogroup 5: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 5: 30 days post dose 2 | 76.4 [66.2 to 84.8] |
  PPAS1: Serogroup 6A: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 6A: 30 days post dose 2 | 88.8 [80.3 to 94.5] |
  PPAS1: Serogroup 6B: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 6B: 30 days post dose 2 | 40.4 [30.2 to 51.4] |
  PPAS1: Serogroup 7F: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 7F: 30 days post dose 2 | 97.8 [92.1 to 99.7] |
  PPAS1: Serogroup 9V: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 9V: 30 days post dose 2 | 88.8 [80.3 to 94.5] |
  PPAS1: Serogroup 14: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 14: 30 days post dose 2 | 96.6 [90.5 to 99.3] |
  PPAS1: Serogroup 18C: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 18C: 30 days post dose 2 | 91.0 [83.1 to 96.0] |
  PPAS1: Serogroup 19A:30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 19A:30 days post dose 2 | 93.3 [85.9 to 97.5] |
  PPAS1: Serogroup 19F: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 19F: 30 days post dose 2 | 98.9 [93.9 to 100] |
  PPAS1: Serogroup 23F: 30 days post dose 2: number analyzed (Participants) | 89 | 0
  PPAS1: Serogroup 23F: 30 days post dose 2 | 71.9 [61.4 to 80.9] |
  PPAS2: Serogroup 1: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 1: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 1: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 1: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 3: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 3: 30 days post dose 3 | 97.8 [92.3 to 99.7] |
  PPAS2: Serogroup 3: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 3: 30 days post dose 4 |  | 92.1 [84.5 to 96.8]
  PPAS2: Serogroup 4: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 4: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 4: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 4: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 5: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 5: 30 days post dose 3 | 98.9 [94.0 to 100] |
  PPAS2: Serogroup 5: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 5: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 6A: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 6A: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 6A: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 6A: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 6B: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 6B: 30 days post dose 3 | 98.9 [94.0 to 100] |
  PPAS2: Serogroup 6B: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 6B: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 7F: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 7F: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 7F: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 7F: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 9V: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 9V: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 9V: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 9V: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 14: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 14: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 14: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 14: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 18C: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 18C: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 18C: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 18C: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 19A: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 19A: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 19A: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 19A: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 19F: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 19F: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 19F: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 19F: 30 days post dose 4 |  | 100 [95.9 to 100]
  PPAS2: Serogroup 23F: 30 days post dose 3: number analyzed (Participants) | 91 | 0
  PPAS2: Serogroup 23F: 30 days post dose 3 | 100 [96.0 to 100] |
  PPAS2: Serogroup 23F: 30 days post dose 4: number analyzed (Participants) | 0 | 89
  PPAS2: Serogroup 23F: 30 days post dose 4 |  | 100 [95.9 to 100]

17. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Measles, Mumps and Rubella (MMR) Antibodies
Description: GMCs of anti-measles and anti-rubella antibodies were measured by bulk IgG enzyme immunoassay (EIA) and anti-mumps antibodies were assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Groups 1, 2 and 3: At 30 days post Dose 3 (12 to 18 MoA); Group 4: At 30 days post Dose 4 (12 to 18 MoA)
Population: PPAS2 was a subset of FAS2. FAS2 included subset of randomized participants who received at least 1 dose of the study vaccine at booster vaccination and had a valid post-booster vaccination blood sample result. Only participants with data collected for each specific serogroup are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 525 | 553 | 94 | 90
Titer
  Anti-measles: 30 days post dose 3: number analyzed (Participants) | 525 | 553 | 94 | 0
  Anti-measles: 30 days post dose 3 | 2780 [2581 to 2995] | 2919 [2739 to 3110] | 3457 [2972 to 4021] |
  Anti-measles: 30 days post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  Anti-measles: 30 days post dose 4 |  |  |  | 3933 [3241 to 4773]
  Anti-mumps: 30 days post dose 3: number analyzed (Participants) | 525 | 553 | 94 | 0
  Anti-mumps: 30 days post dose 3 | 83.3 [77.5 to 89.6] | 86.1 [80.5 to 92.1] | 105 [90.4 to 121] |
  Anti-mumps: 30 days post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  Anti-mumps: 30 days post dose 4 |  |  |  | 121 [105 to 141]
  Anti-rubella: 30 days post dose 3: number analyzed (Participants) | 525 | 553 | 94 | 0
  Anti-rubella: 30 days post dose 3 | 56.8 [53.2 to 60.6] | 56.0 [52.5 to 59.8] | 72.8 [62.7 to 84.6] |
  Anti-rubella: 30 days post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  Anti-rubella: 30 days post dose 4 |  |  |  | 74.4 [63.7 to 86.7]

18. Secondary Outcome: Percentage of Participants Who Achieved Vaccine Response for Measles, Mumps and Rubella (MMR) Antibodies
Description: GMCs of anti-measles and anti-rubella antibodies were measured by bulk IgG EIA and anti-mumps antibodies were assessed by ELISA. Vaccine response against anti-measles, anti-mumps, anti-rubella antibodies were defined as percentage of participants with anti-measles, anti-mumps, anti-rubella antibody concentration that met the respective mentioned criterion: measles: >=255 mIU/mL; mumps: >=10 mumps antibody units/mL and rubella: >=10 IU/mL. Percentages are rounded off to the tenth decimal place.
Time Frame: Groups 1, 2 and 3: At 30 days post Dose 3 (12 to 18 MoA); Group 4: At 30 days post Dose 4 (12 to 18 MoA)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
Number analyzed (Participants) | 525 | 553 | 94 | 90
Percentage of participants
  Anti-measles: 30 days post dose 3: number analyzed (Participants) | 525 | 553 | 94 | 0
  Anti-measles: 30 days post dose 3 | 98.3 [96.8 to 99.2] | 99.1 [97.9 to 99.7] | 100 [96.2 to 100] |
  Anti-measles: 30 days post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  Anti-measles: 30 days post dose 4 |  |  |  | 97.8 [92.2 to 99.7]
  Anti-mumps: 30 days post dose 3: number analyzed (Participants) | 525 | 553 | 94 | 0
  Anti-mumps: 30 days post dose 3 | 98.7 [97.3 to 99.5] | 98.7 [97.4 to 99.5] | 100 [96.2 to 100] |
  Anti-mumps: 30 days post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  Anti-mumps: 30 days post dose 4 |  |  |  | 100 [96.0 to 100]
  Anti-rubella: 30 days post dose 3: number analyzed (Participants) | 525 | 553 | 94 | 0
  Anti-rubella: 30 days post dose 3 | 98.7 [97.3 to 99.5] | 97.3 [95.6 to 98.5] | 98.9 [94.2 to 100] |
  Anti-rubella: 30 days post dose 4: number analyzed (Participants) | 0 | 0 | 0 | 90
  Anti-rubella: 30 days post dose 4 |  |  |  | 100 [96.0 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs), serious adverse events (SAEs) and all-cause mortality (deaths) were collected from the study vaccine administration (Day 0) until 30 days after the last vaccination (Visit 5 [13 to 19 MoA] for Groups 1, 2, and 3 and Visit 6 [13 to 19 MoA] for Group 4), up to 14 to 20 MoA.
Description: Analysis was performed on the safety analysis set (SafAS)which included those participants who had received at least 1 dose of the study vaccine(s) and had any safety data available.
Arm/Group | Group 1: MenACYW | Group 2: Nimenrix | Group 3: MenACYW | Group 4: MenACYW
All-Cause Mortality (participants affected / at risk) | 0/696 | 0/706 | 0/112 | 0/108
Serious Adverse Events (participants affected / at risk) | 51/696 | 57/706 | 8/112 | 3/108
Other Adverse Events (participants affected / at risk) | 678/696 | 680/706 | 107/112 | 103/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW (N=696) | Group 2: Nimenrix (N=706) | Group 3: MenACYW (N=112) | Group 4: MenACYW (N=108)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital Hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphatic Malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Food Protein-Induced Enterocolitis Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 6 (7) | 5 (5) | 0 (0) | 0 (0)
Bronchitis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exanthema Subitum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Gastroenteritis Adenovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 2 (6) | 2 (2) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 2 (2)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns Third Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exposure To Toxic Agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight Gain Poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Testicular Yolk Sac Tumour Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clinically Isolated Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Petit Mal Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Respiration Abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW (N=696) | Group 2: Nimenrix (N=706) | Group 3: MenACYW (N=112) | Group 4: MenACYW (N=108)
Diarrhoea (Gastrointestinal disorders) | 55 (63) | 37 (44) | 4 (4) | 2 (2)
Teething (Gastrointestinal disorders) | 99 (142) | 93 (135) | 7 (10) | 15 (28)
Toothache (Gastrointestinal disorders) | 13 (16) | 8 (13) | 6 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 196 (268) | 197 (271) | 25 (32) | 27 (33)
Crying (General disorders) | 579 (1274) | 579 (1279) | 74 (138) | 75 (158)
Injection Site Bruising (General disorders) | 110 (194) | 124 (188) | 3 (5) | 4 (7)
Injection Site Erythema (General disorders) | 537 (2207) | 520 (2169) | 61 (173) | 58 (188)
Injection Site Haematoma (General disorders) | 55 (97) | 56 (92) | 7 (10) | 16 (21)
Injection Site Induration (General disorders) | 68 (137) | 52 (91) | 6 (8) | 4 (6)
Injection Site Mass (General disorders) | 64 (139) | 60 (134) | 3 (3) | 1 (1)
Injection Site Pain (General disorders) | 562 (2842) | 566 (2851) | 88 (430) | 76 (450)
Injection Site Swelling (General disorders) | 422 (1445) | 417 (1458) | 41 (118) | 47 (164)
Pyrexia (General disorders) | 375 (570) | 345 (537) | 46 (57) | 42 (70)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 11 (12) | 12 (13)
Conjunctivitis (Infections and infestations) | 16 (16) | 21 (21) | 4 (4) | 7 (9)
Gastroenteritis (Infections and infestations) | 10 (10) | 18 (18) | 6 (6) | 9 (11)
Nasopharyngitis (Infections and infestations) | 65 (80) | 64 (76) | 2 (2) | 8 (8)
Respiratory Tract Infection (Infections and infestations) | 7 (8) | 12 (13) | 7 (7) | 2 (2)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1) | 18 (21) | 22 (31)
Rhinitis (Infections and infestations) | 47 (56) | 47 (50) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 54 (64) | 61 (71) | 3 (3) | 5 (6)
Decreased Appetite (Metabolism and nutrition disorders) | 389 (594) | 372 (566) | 60 (90) | 58 (103)
Somnolence (Nervous system disorders) | 529 (1094) | 545 (1060) | 67 (112) | 75 (155)
Irritability (Psychiatric disorders) | 600 (1413) | 608 (1426) | 91 (190) | 86 (217)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (4) | 6 (7)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (4) | 6 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 16 (18) | 23 (25) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT03547271/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT03547271/SAP_001.pdf